| 1 | CLINICAL RESEARCH PROTOCOL | |
|---|---|---|
| 1 2 3 | NATIONAL INSTITUTE OF DIABETES AND DIGESTIVE AND KIDNEY DISEASES | |
| 4<br>5<br>6 | DATE: August 3, 2016 CLINICAL PROTOCOL NO.: 15-DK-0082 | |
| 7<br>8<br>9 | IND NO: xx,xxx<br>IND Name: xx<br>IND HOLDER: | |
| 10<br>11 | TITLE: Mechanisms Associated with Favorable Response to Peginterferon-Alpha Add-on | Therapy |
| 12 | Following Long-term Nucleos(t)ide Analogue Treatment in Patients with Chronic Hepatiti | s B |
| 13 | SHORT TITLE: Add on PegIFN to NUC Therapy for CHB | |
| 14<br>15<br>16<br>17 | <b>IDENTIFYING WORDS</b> : Peginterferon alfa-2a Nucleos(t)ide analogues, Chronic Hepatitis Biopsy, HBeAg loss, HBsAg loss, Interferon stimulating gene. | B, Liver |
| 18<br>19<br>20 | <b>PRINCIPAL INVESTIGATOR</b> : Marc Ghany, M.D., MHSc, Liver Diseases Branch (LDB), Nation Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)* | onal |
| 21<br>22<br>23<br>24 | ASSOCIATE SENIOR INVESTIGATORS: T Jake Liang, Chief, Liver Diseases Branch (LDB), National Institute of Diabetes and Digest Kidney Diseases (NIDDK)* Barbara Rehermann, M.D., Senior Investigator, LDB, NIDDK | ive and |
| 25<br>26<br>27<br>28<br>29 | Edward Doo, M.D., LDRB, Division of Digestive Diseases and Nutrition, NIDDK* Theo Heller, M.D., Investigator, LDB, NIDDK* Yaron Rotman, M.D. Investigator, LDB, NIDDK* Christopher Koh, M.D. Staff Physician, LDB, NIDDK* Elizabeth Wright, Ph.D. OD, NIDDK | |
| 30<br>31 | David Kleiner, M.D., PhD., Laboratory of Clinical Pathology, NCI | |
| 32<br>33<br>34<br>35<br>36<br>37<br>38 | ASSOCIATE STAFF INVESTIGATORS: Ahmad Alawad, M.D. Medical Staff Fellow, LDB, NIDDK* Devika Kapuria, M.D. Medical Staff Fellow, LDB, NIDDK* Gil Ben-Yakov, M.D., Medical Staff Fellow, LDB, NIDDK* Elenita Rivera, R.N., Research Nurse, LDB, NIDDK Amy Huang R.N. Research Nurse, LDB, NIDDK | |
| 39<br>40<br>41 | Non-NIH Investigators<br>Gavin Cloherty, PhD, Abbott Diagnostics | |
| 42<br>43 | *Investigators with this designation will obtain informed consent for this protocol. | |
| 44<br>45<br>46<br>47 | <b>ESTIMATED DURATION OF STUDY</b> : 3 Years <b>NUMBER AND TYPE OF PATIENTS</b> : 60 patients with chronic hepatitis B, ages above 18 y male and female | ears, both |
| 48<br>49<br>50 | SUBJECTS OF STUDY: Number of patients: 60 Sex: Male & Female Volunteers: None Age Range: Above 18 years | |
| 51<br>52<br>53 | <b>PROJECT USES IONIZING RADIATION</b> : Yes, for medical indications only. | |
| 53<br>54 | PROJECT USES "DURABLE POWER OF ATTORNEY": No | |

| 1<br>2<br>3 | OFF-SITE PROJECT: No | MULTI-INSTITUTIONAL PROJECT: No |
|-------------|----------------------|---------------------------------|
| 4 | | |
| 5 | | |
| 6 | | |
| 7 | | |

1 Précis

2

4

5

6

7

8

9

10

11

12

13

14

15

16

17

18

19

20

21

22

23

24

25

26

27

28

Chronic hepatitis B virus (HBV) infection is a leading cause of liver associated morbidity and mortality. Currently available first-line therapies for treatment of chronic hepatitis B include pegylated interferon-alpha and the nucleos(t)ide analogues (NUCs) entecavir and tenofovir. These were shown to effectively suppress viral replication, but their ability to induce durable off-treatment response is limited to a small subset of patients. Combination treatment with peginterferon and NUCs has been attempted in several randomized controlled trials, with no apparent advantage over either agent given alone. In these studies however, treatment with peginterferon was initiated either simultaneously or shortly after NUCs administration. The efficacy of peginterferon following longterm viral suppression with NUCs was only tested in one small pilot study, nevertheless showing 60% HBsAg loss rate. The underlying mechanisms responsible for improved efficacy of peginterferon in this setting are unknown and warrant further investigation. In this single arm study we propose to evaluate the efficacy and mechanisms associated with response to peginterferon add-on therapy following a minimum of 192 weeks of viral suppression induced by NUCs in a group of chronic HBV infected patients. Sixty patients with either HBeAg positive (n=30) or negative (n=30) chronic HBV infection will be enrolled to this study. After medical evaluation and pretreatment liver biopsy, treatment with subcutaneous injections of pegylated interferon alpha-2a 180 µg per week will be given for a total of 24 weeks, followed by an off-treatment evaluation period of 48 weeks. A second liver biopsy will be performed six hours following the first peginterferon injection. Primary end-point for this study will be the change in interferon-stimulated-genes response before and after first interferon injection in responders versus non-responders to treatment. The responsiveness to IFN-based therapy of treatment responders vs nonresponders will additionally be evaluated by studying intrahepatic and peripheral blood natural killer cells. The study will also assess HBeAg and HBsAg loss and seroconversion rates in comparison to historical controls treated with either peginterferon or NUCs monotherapy. Finally, we will assess whether treatment responders develop an HBV-specific T cell response similar in quantity and quality to that of patients who spontaneously resolve HBV infection.

| 1 | Table of Contents | |
|---|---|---|
| 2 | Précis | 3 |
| 3 | BACKGROUND | 5 |
| 4 | HYPOTHESIS | 8 |
| 5 | SPECIFIC AIMS | 8 |
| 6 | PROTOCOL OVERVIEW | |
| 7 | INCLUSION/EXCLUSION CRITERIA | |
| 8 | Inclusion criteria: HBeAg positive group | 9 |
| 9<br>10 | Inclusion criteria: HBeAg negative group<br>Exclusion criteria (for both eAg positive and negative patients) | |
| 11<br>12 | STUDY DESIGN AND PROCEDURESScreening | |
| 13 | Admission for pretreatment liver biopsy | 12 |
| 14<br>15 | Initiation of Treatment | |
| 16 | On-treatment liver biopsy | |
| 17 | Table 1: List of study related procedures | |
| 18 | ASSESSMENT OF RESPONSE | 18 |
| 19 | Clinical Definitions | |
| 20<br>21 | Primary end-pointSecondary endpoints | |
| 22 | DOSE CHANGES | |
| 23 | Stopping peginterferon therapy: | |
| 24 | Stopping NUCs therapy | |
| 25<br>26 | Peginterferon Dose Modifications | |
| 27 | STATISTICAL ANALYSIS | |
| 28 | Power calculation | |
| 29 | Demographics and Baseline Characteristics | |
| 30<br>31 | Analysis planAnalysis methodology | |
| 32 | HAZARDS AND DISCOMFORTS | |
| 33 | RISK IN RELATION TO BENEFIT | |
| 34 | ADVERSE EVENT REPORTING | |
| 35 | DATA AND SAFETY MONITORING | |
| 36 | CLINICAL MONITORING PLAN | |
| 37 | ENROLLMENT OF CHILDREN, WOMEN AND MINORITY INDIVIDUALS | |
| 38 | RESEARCH USE, STORAGE AND DISPOSITION OF HUMAN SAMPLES AND DATA | |
| 39 | RECRUITMENT PLAN | |
| 40 | CONSENT PROCESS | |
| 41 | COMPENSATION | |
| 42 | REFERENCES | |
| 43<br>44 | RLI ERLINGES | 34 |

#### BACKGROUND

345

6

7

8

9

10

2

It is estimated that there are over 350 million persons with chronic hepatitis B virus (HBV) infection worldwide [1] Globally, chronic HBV infection is the leading cause of cirrhosis and hepatocellular carcinoma accounting for  $\sim$ 620,000 deaths annually [2] Epidemiological studies have demonstrated a strong association between high viral levels and worse outcome of chronic HBV infection [3, 4]. Thus, the goal of therapy is long-term, sustained suppression of HBV replication. Current first line recommendations for treatment of chronic HBV infection include entecavir, tenofovir (nucleos(t)ide analogues) or peginterferon-alpha [1, 5, 6].

111213

14

15

16

17

18

19

20

21

22

23

24

25

26

27

28

29

30

31

32

33

34

35

36

NUCs with potent activity against the HBV reverse transcriptase and high barrier to resistance have been very effective at suppressing viral replication and were shown to be associated with improved clinical outcomes including reversal of cirrhosis [7, 8]. However, discontinuing therapy after one year is associated with high relapse rates and therefore most patients require long-term therapy to maintain suppression of viral replication [9-11]. Even with long-term use of NUCs, only about 50% of persons who were initially HBeAg positive undergo HBeAg seroconversion (the endpoint of therapy for HBeAg positive persons) [12, 13] and among those who were initially HBeAg negative, only about 1%-2% experience HBsAg seroconversion (the endpoint of therapy for HBeAg negative persons) [14, 15] Unfortunately, there are substantial costs associated with long-term therapy and there is the potential for serious side effects including renal toxicity and possibly loss of bone mass [16-20] Thus, new agents or approaches are needed to manage patients with chronic HBV infection. One approach that has been taken to improve HBsAg loss was to combine the two most potent NUCs. In one notable trial, the efficacy and safety of entecavir monotherapy was compared to the combination of entecavir and tenofovir in persons with HBeAg positive and negative chronic HBV infection. After 96 weeks of therapy, a comparable proportion of patients in each study arm achieved the primary end point of a level of HBV DNA<50 IU/mL (83.2% vs 76.4%, respectively), indicating no benefit of a combination NUC approach over potent monotherapy [21]. Another approach was to combine a nucleoside analogue with peginterferon. This strategy is theoretically appealing as the combined effect of peginterferon, an immunomodulator, and a nucleos(t)ide analogue, a potent inhibitor of viral replication, may result in a synergistic anti-viral effect. However, several trials comparing the efficacy of combination peginterferon-NUCs therapy to either agent alone failed to show a clear advantage of combination therapy over either agent alone. Four randomized controlled trials comparing peginterferon alfa and NUCs (either lamivudine or adefovir) to peginterferon alone or NUCs alone have been conducted in persons with HBeAg positive and negative chronic HBV infection. [22-25]. All studies reported greater on-treatment viral suppression with the combination regimen compared to either agent alone, but higher rates of sustained off-treatment viral suppression with the combination regimen were only achieved in comparisoin to NUCs alone but not to peginterferon alone. Thus, there is really no advantage of combination peginterferon and lamivudine or adefovir to peginterferon alone, when treatment with the two agents is initiated simultaneously.

Studies assessing baseline predictors of response to peginterferon have shown that high viral levels are associated with a less favorable response in both HBeAg positive and negative HBV infected patients [26, 27]. In this context, it may be postulated that high viral titers may inhibit the action of peginterferon and that combination peginterferon plus a nucleos(t)ide analogue may be more effective if the peginterferon is preceded by a lead-in period of the nucleos(t)ide analogue. In one study testing this strategy, 185 persons with HBeAg positive chronic hepatitis B were randomized to receive either entecavir monotherapy for 48 weeks or a lead-in period of 24 weeks of entecavir followed by 24 weeks of combination entecavir plus peginterferon [28]. At end-of-treatment more patients in the combination arm, 19%, achieved the primary endpoint of HBeAg seroconversion compared to the entecavir monotherapy arm, 10%. This difference however was not statistically significant (p=0.095), and there was no peginterferon monotherapy arm. However, in a prespecified multivariate analysis adjusted for differences in HBV DNA at the start of the randomized therapy phase, add-on peginterferon was significantly associated with a 4.78-fold increase in response rate (P = .004). It is possible though that a longer period of viral suppression is required to improve the efficacy of peginterferon therapy in combination with a NUCs. Indeed in a small pilot study in which peginterferon was added after a minimum period of 3 years of entecavir therapy with complete viral suppression, showed that 60% of persons developed HBsAg loss [29]. These provocative results suggest that a peginterferon add-on strategy following a substantial period of nucleos(t)ide induced viral suppression, may result in high rates of HBsAg seroconversion. The underlying mechanisms responsible for improved efficacy of peginterferon in this setting, are unknown, or for that matter the mechanism of action of peginterferon in chronic HBV infection and warrant further investigation.

IFN- $\alpha$  is a naturally occurring cytokine with broad anti-viral activity. Its anti-viral effect is mediated through induction of a diverse set of target genes, referred to as IFN-stimulated genes (ISGs)[30]. This results in inhibition of HBV replication through a variety of mechanisms including a block of RNA-containing core particle formation, an accelerated decay of replication-competent core particles, and degradation of the pre-genomic RNA [31-33]. Recently, IFN- $\alpha$  was also shown to inhibit HBV replication by decreasing RNA transcription from cccDNA. This effect was mediated through epigenetic repression of cccDNA (via histone hypoacetylation), as well as by active recruitment to the cccDNA of transcriptional co-repressors [34].

In addition to its direct anti-viral activity, IFN- $\alpha$  is also a potent immunomodulator with robust effects on cells of the innate immune system, such as natural killer cells (NK). NK cells consistitute the largest lymphocyte population in the liver and can exert antiviral function via direct cytotoxic mechanisms and via indirect cytokine (e.g. IFN-gamma mediated) mechanisms. NK cells respond to IFN-a and we have previously shown that the response of peripheral blood NK cells to Peg-interferon correlates well with the overal response and clinical outcome of PegIFN-based regimens in chronic HCV infection [35, 36]. Interferon also modulates the adaptive, T cell-mediated response. T cells are typically impaired in their antiviral function in chronic HBV infection. This impairment has been attributed to upregulation of inhibitory molecules such as PD-1, Tim-3, CTLA-4 and others due to chronic T cell receptor stimulation by HBV antigens resulting in downregulation of virus-specific T cell response of infected patients [37]. In this protocol we will determine whether a decrease in HBV titer by NUCs improves the innate and adaptive immune response to PegIFN. We postulate that in patients with chronic HBV infection, who have long-term viral suppression due to NUCs therapy, the addition of peginterferon will lead to HBeAg or HBsAg seroconversion. We plan to explore the clinical response and possible mechanisms involved during therapy with peginterferon alfa when added to long-term nucleoside therapy in patients with chronic HBV infection (both HBeAg-positive and -negative). We hypothesize that the extended pretreatment with NUCs will modify the responsiveness to peginterferon. These effects will be studied by analyzing the expression pattern of ISGs, the response of NK cells prior to and after peginterferon injection resulting in improved transcriptional control of cccDNA, the induction of antibodies against HBe and HBsAg and T cell responses. Primary endpoints of this trial will be the changes in expression levels of ISG's, intrahepatic total HBV DNA and cccDNA content, changes in NK cell effector cell function measured before and following a single dose of peginterferon stratified by treatment response and the rates of HBeAg and HBsAg loss and seroconversion in HBeAg positive patients, HBsAg loss and seroconversion rate in HBeAg negative patients. Secondary endpoints will be the induction of HBV-specific memory T cell responses. A post-hoc analysis will stratify reponse rates upon available viral genotype data and duration of NUC therapy prior to study enrollment. Other secondary end-points will include changes in quantitative HBeAg and HBsAg levels during therapy and safety of the combination regimen. Serological response rates, qHBsAg kinetics and safety end-points will be compared to historical controls of published multicenter randomized trials comparing the efficacy of peginterferon and

3334

1

2

3

4

5

6

7

8

9

10

11

12

1314

15

16

17

18

19

20

21

22

23

24

25

26

27

28

29

30

31

32

NUCs in eAg positive and negative HBV carriers

1 HYPOTHESIS

In patients with chronic hepatitis B infection, under long-term viral suppression maintained by NUCs treatment, peginterferon add-on therapy will result in a greater proportion of subjects achieving serological response compared to before peginterferon was added. We hypothesize that response to treatment will be accompanied by measurable changes in host-response gene transcription profile, immune cell activation and function, and quantitative viral biomarker levels.

U

## 9 SPECIFIC AIMS

- 1. To assess the changes in ISG profile and NK cell function after a single dose of peginterferon in patients receiving long-term NUCs with maintained viral suppression
- 2. To determine rates of HBeAg and HBsAg loss with or without seroconversion and induction of HBV-specific memory T cells to peginterferon add-on treatment in eAg positive and negative HBV carriers on long-term NUC treatment.
- 3. To identify pre- and on-treatment predictors of serological response to peginterferon add-on/nucleos(t)ide combination therapy.
- 4. To determine if there are differences in epigenetic regulation of cccDNA between HBeAg positive and negative CHB at baseline and following a single dose of peginterferon treatment

# 21 PROTOCOL OVERVIEW

We intend to enroll a total of 60 patients with HBeAg positive (n=30) and HBeAg negative (n=30) chronic HBV infection, who have been on-treatment with one or more nucleos(t)ide analogues for at least 192 weeks prior to study enrollment with maintained viral suppression (HBV DNA level <100 IU/ml). After a thorough medical evaluation and liver biopsy, participants will receive therapy with subcutaneous injections of peginterferon-alpha 2a at a dose of 180mcg per week for a total of 24 weeks. A second liver biopsy will be performed 6 hours following the first peginterferon injection for the purpose of assessing ISGs, intrahepatic NK cell quantity and function and intrahepatic viral biomarker response patterns. Most interferon induced genes achieve maximal response in the liver and periphery within 4 hours, begin to decline by 8 hours, and return to baseline levels by 24 hours post-administration of interferon. Because peginterferon is slower to be absorbed we have selected the six hour rather that a four hour time point.[38]

| 1 | Patient | s will be followed carefully on weeks 0, 2, 4, 8, 12 and 24 during treatment and at 12 week |
|---|---|---|
| 2 | interva | ls thereafter until 48 weeks post-treatment. |
| 3 | During | study visits patients will be assessed for compliance with study medications, as well as the |
| 4 | develop | development of any treatment related side effects and/or adverse reactions. In addition, blood will |
| 5 | be drav | vn periodically for the assessment of routine blood tests, quantitative viral biomarker levels, |
| 6 | serolog | ical response markers and immune cell functional status. |
| 7 | | |
| 8<br>9 | | INCLUSION/EXCLUSION CRITERIA |
| 10<br>11 | Inclusi | on criteria: HBeAg positive group |
| 12 | 1) | Age >18 years and older, male or female. |
| 13 | 2) | Known serum HBsAg and HBeAg positivity at the time of screening. |
| 14 | 3) | Ongoing treatment with one or more NUCs for at least 192 weeks before study entry. |
| 15 | | Subjects may have a brief interruption of treatment for medical reasons (e.g. breast feeding) |
| 16 | | not to exceed 8 weeks and none within the 48 weeks before study entry. |
| 17 | 4) | HBV DNA levels <100 IU/mL, measured at least 12 months prior to, and upon enrollment to |
| 18 | | the study. |
| 19 | 5) | ALT level ≤2 ULN based on at least two determinations taken at least one month apart |
| 20 | | during the 24 weeks before study entry with the second being at time of screening |
| 21 | 6) | Written informed consent |
| 22 | | |
| 23<br>24 | Inclus | ion criteria: HBeAg negative group |
| 25 | 1) | Age >18 years and older, male or female. |
| 26 | 2) | Known serum HBsAg positivity and HBeAg negativity at the time of screening. |
| 27 | 3) | Ongoing treatment with one or more NUCs for at least 192 weeks before study entry. |
| 28 | | Subjects may have a brief interruption of treatment for medical reasons (e.g. breast feeding) |
| 29 | | not to exceed 8 weeks and none within the 48 weeks before study entry. |
| 30 | 4) | HBV DNA levels $<$ 100 IU/mL, measured at least 12 months prior to, and upon enrollment to |
| 31 | | the study |
| 32 | 5) | ALT level ≤2 ULN based on at least two determinations taken at least one month apart |
| 33 | | during the 24 weeks before study entry with the second being at time of screening |
| 34 | 6) | Written informed consent |
| 35 | | |

#### 1 Exclusion criteria (for both eAg positive and negative patients) 2 3 1) Co-infection with HDV as defined by the presence of anti-HDV in serum and/or HDV antigen 4 in the liver. 5 2) Co-infection with HCV as defined by the presence of HCV RNA in serum. 6 3) Co-infection with HIV as defined by the presence of anti-HIV in serum. 7 4) Decompensated liver disease as defined by serum bilirubin >2.5 mg/dL (with direct bilirubin 8 > 0.5 mg/dL), prothrombin time of greater than 2 seconds prolonged, a serum albumin of 9 less than 3 g/dL, or a history of ascites, variceal bleeding or hepatic encephalopathy. 10 5) Presence of other causes of liver disease, (i.e. hemochromatosis, Wilson disease, alcoholic 11 liver disease, severe nonalcoholic steatohepatitis defined as the presence of marked 12 ballooning injury on liver biopsy, alpha-1-anti-trypsin deficiency). 13 6) A history of organ transplantation or in the absence of organ transplantation, any 14 immunosuppressive therapy requiring the use of more than 5 mg of prednisone (or its 15 equivalent) daily. 16 7) Significant systemic illness other than liver diseases including congestive heart failure, renal 17 failure, chronic pancreatitis and diabetes mellitus with poor control, that in the opinion of 18 the investigator may interfere with therapy. 19 8) Pregnancy or inability to practice contraception in patients capable of bearing or fathering 20 children 21 9) Lactating women. 22 10) Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver 23 that is suggestive of HCC, or an alpha-fetoprotein level of greater than 500 ng/mL. 24 11) eGFR < 50 ml/min, serum creatinine > 1.3 mg/dl or urine protein >1 gram/24-hours 25 12) History of hypersensitivity to pegylated interferon-alpha 26 13) Platelet count < 70 mm<sup>3</sup>/dL 27 14) Hgb <12 g/dL for males and <11 g/dL for females 28 15) Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, 29 bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, 30 in the investigator's opinion, might interfere with participation in the study. 31 16) History of malignancy or treatment for a malignancy within the past 3 years (except 32 adequately treated carcinoma in situ or basal cell carcinoma of the skin). 33 17) Any medical condition requiring, or likely to require, chronic systemic administration of 34 corticosteroids or other immunosuppressive medications during the course of this study.

18) History of immune-mediated disease, or cerebrovascular, chronic pulmonary or cardiac

disease associated with functional limitation, retinopathy, uncontrolled thyroid disease,

35

| 1 | poorly controlled diabetes or uncontrolled seizure disorder, as determined by a study |
|---|---|
| 2 | physician. |
| 3 | 19) Presence of conditions that, in the opinion of the investigators, would not allow the patient |
| 4 | to be followed in the current study for at 1 year. |
| 5 | 20) For subjects who interrupt therapy, documentation of a viral load >1,000 IU/ml while off |
| 6 | therapy. |
| 7 | |
| 8 | STUDY DESIGN AND PROCEDURES |
| l0<br>l1 | Screening |
| 2 | Eligible patients will be seen in the outpatient liver clinic of the NIH Clinical Center. At the screening |
| 13 | visit, potential benefits and risks associated with the study will be explained to the study participant: |
| 4 | by an investigator in laymen's language. Written informed consent will be obtained and documented |
| 15 | in the participant's chart. Whenever possible, the informed consent form will be provided to the |
| 16 | potential participants in advance. Only the principal and associate investigators from the Liver |
| 17 | Disease Branch, NIDDK, will be eligible to obtain consent for this study. |
| 18 | |
| 9 | The following screening procedures will be performed: |
| 20 | (1) Obtain signed informed consent |
| 21 | (2) History and physical examination |
| 22 | (3) Symptom questionnaire |
| 23 | (4) Fatigue questionnaire (Promise 7) |
| 24 | (5) Visual analogue scale |
| 25 | (6) Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, |
| 26 | phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, |
| 27 | LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC |
| 28 | (hematocrit, hemoglobin, white blood cell count and differential, platelet count). |
| 29 | Testing will also be done for anti-HAV, HBsAg, anti-HBs, HBeAg, anti-HBe, anti-HBc, |
| 30 | anti-HCV, and stored sample for IL-28b testing. Baseline HBV DNA level by quantitativ |
| 31 | PCR (COBAS Ampliprep/COBAS Taqman HBV v2.0 Test: Roche Diagnostics, lower limit |
| 32 | of quantification 116 copies /ml or 20 IU/ml, lower limit of detection 6 IU/ml) |
| 33 | (7) Extended blood panel: alpha fetoprotein, gGT, immunoglobulins, rheumatoid factor, |
| 34 | ANUCs, SMA, lipid panel, thyroid panel, INR, reticulocyte count, ESR. |

| 1 | (8) Research blood- one 10 ml serum and one 10 ml plasma tube stored frozen in 0.5-1.0 |
|---|---|
| 2 | mL aliquots). The stored serum and plasma will be used to measure selected cytokines, |
| 3 | interferon-stimulated gene products [including IP10], quantitative HBsAg level (by |
| 4 | using the Roche Elecsys HBsAg automated quant assay) and for future research. |
| 5 | (9) Fifty milliliters of whole blood (green top tubes) for baseline immunological studies: NK |
| 6 | cell responses, CD4+ and CD8+ T cell HBV specific responses (peripheral blood |
| 7 | mononuclear cell [PBMC] studies) |
| 8 | (10) Urine tests: routine urinalysis and a pregnancy test for females of childbearing |
| 9 | notential |

(11) Transient elastography

1011

#### Admission for pretreatment liver biopsy

12 13 14

15

16

17

18

19

20

21

22

23

24

25

26

27

28

29

30

labs, they will have 12 weeks to complete the liver biopsy and to begin add-on therapy with peginterferon. Eligible patients will be admitted to 5NW to undergo a percutaneous liver biopsy. The initial liver biopsy will be mostly for research purposes to measuring baseline levels of ISG expression, pregenomic and cccDNA concentration and frequency and activity of liver infiltrating HBV-specific NK cells but will also be used for the purpose of grading and staging of liver disease before treatment and will provide useful information to the clinician and patient on whether the liver disease is improving on current therapy. Grading and staging of the liver biopsy will performed by an expert hepatopathologist blinded to the clinical information using the modified Ishak scoring system. This includes the histological activity index (HAI) for inflammation and necrosis (scores ranging from 0 to 18). Fibrosis will be staged using the Ishak scoring system (0-6, 0=no fibrosis, 6=cirrhosis). Slides will also be immunostained for HBsAg, HBcAg, and HDV antigen by peroxidase-antiperoxidase techniques and scored as 0, 1, 2 or 3+ based upon the percent of cells reactive for each viral antigen (0=none, 1=10%, 2=11% to 50% and 3=≥51% of hepatocytes). Liver-infiltrating lymphocytes will be assessed for frequency and function of NK cells. m-RNA levels of ISG's, immune cell markers and chemokines/cytokines will be quantitated by real-time PCR or nanostring. Intrahepatic pregenomic and cccDNA will also be quantitated by Southern

Once patients are deemed eligible to participate in the study based on results of the screeing

31 32

> 33 34

35

36

The following will be obtained on admission:

1) Brief clinical evaluation

blotting or real-time PCR.

2) Review patient's eligibility for study

| 2 | 4) | Visual analogue scale |
|---|---|---|
| 3 | 5) | Fatigue questionnaire (Promise 7) |
| 4 | 6) | Abdominal ultrasound, CXR and 12 lead ECG (if not done within previous 6 months) |
| 5 | 7) | Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, |
| 6 | | glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline |
| 7 | | Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin |
| 8 | | white blood cell count and differential, platelet count). |
| 9 | 8) | HBV DNA viral load, qualitative and quantitative HBeAg and HBsAg measurement |
| 10 | 9) | 50 mL of blood in heparinized green top tubes for NK and T cell analysis. |
| <ul><li>11</li><li>12</li></ul> | 10) | Blood sample for storage (5 mL of blood separated into serum and stored frozen in 0.5-1.0 mL aliquots) |
| 13 | 11) | Liver biopsy cut into four sections, one (at least 1.5 cm) placed in formalin for routine light |
| 14 | | microscopy and the other 3 (.3cm, .5cm and 1 cm) placed in RNA later and flash frozen in |
| 15 | | liquid nitrogen 24 hours later for RNA and protein analyses and flow cytometry. A liver |
| 16 | | biopsy fragment of > 5 mm will be used to assess the frequency and function of NK cells. |
| 17 | 12) | Discharge from hospital |
| 18 | | |
| 19 | | |
| 20<br>21 | Initiati | on of Treatment |
| 22 | Patient | s will be stratified on the basis of HBeAg status into 2 groups of 30 patients each, to receive |
| 23 | peginte | rferon-alpha 2a (PEGASYS®, Roche), 180 mcg per week administered by subcutaneous |
| 24 | injectio | n for a total of 24 weeks. Patients will continue treatment with their previous nucleosi(t)ide |
| 25 | analogu | ne regimen during the treatment and follow-up phases of this study. |
| 26 | Patient | s will be seen in the outpatient clinic at weeks 2, 4, 8, 12, and 24, during treatment phase, at |
| 27 | 12 wee | k intervals thereafter up to 48 weeks post-therapy |
| 28 | Compli | ance will be monitored by medication diaries and counting of the residual vials returned at |
| 29 | outpati | ent visits. The side effects will be monitored regularly at each visit during the treatment phase |
| 30 | of the s | tudy by symptom questionnaires. Peginterferon alfa-2a will be dose reduced or stopped per |
| 31 | the dos | e reduction and stopping rules for peginterferon alfa-2a. Peginterferon alfa-2a treatment can |
| 32<br>33 | be resta | arted if the adverse event resolves and the patient is willing to re-start the medication. |
| 34<br>35 | On-trea | atment liver biopsy |

3) Symptom questionnaire

| 1 | At day 0, all patients will be readmitted to the NIH Clinical Center to start therapy with peginterfer | on |
|---|---|---|
| 2 | alfa-2a and to undergo a repeat liver biopsy. Biopsy will be scheduled at 6 hours following the first | t |
| 3 | injection of peginterferon, for the purpose of assessing ISG response pattern following the initial | |
| 4 | exposure to peginterferon. Liver tissue will also be subjected to routine histopathological grading | |
| 5 | and staging as well as for immune cell, quantitative viral kinetic and cccDNA epigenetic studies as | |
| 6 | previously described. | |
| 7 | | |
| 8 | Since the hypothesis to be tested in this study is that response to treatment peginterferon (i.e. loss | of |
| 9 | HBeAg and HBsAg or both) is mediated by changes in hepatocyte gene transcription profile, it is | |
| 10 | necessary to obtain liver tissue at two time points-before and 6 hours after the first dose of | |
| 11 | interferon. Performing two liver biopsies within 12 weeks or even as short as 24 hours has been | |
| 12 | performed in other Liver Disease Branch studies and has not been associated with an increase in t | he |
| 13 | complication rate or lower patient acceptance. | |
| 14 | | |
| 15 | | |
| 16 | Monitoring | |
| 17 | Monitoring | |
| 18 | <u>Day 0</u> | |
| 19 | | |
| 20 | 1) Brief clinical evaluation | |
| 21 | 2) Review patient's eligibility for study | |
| 22 | 3) Symptom questionnaire | |
| 23 | 4) Visual analogue scale | |
| 24 | 5) Fatigue questionnaire (Promise 7) | |
| 25 | 6) Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, | |
| 26 | glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline | |
| 27 | Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglo | oin, |
| 28 | white blood cell count and differential, platelet count). | |
| 29 | 7) Females of child bearing potential: Pregnancy test | |
| 30 | 8) HBV DNA, qualitative and quantitative HBeAg, HBsAg, measurements | |
| 31 | 9) 30 mL of blood in heparinized green top tubes for NK and T cell analysis prior to PegIFN | |
| 32 | injection and 30 mL of blood in heparinized green top tubes for NK and T cell analysis 6h | |
| 33 | after PegIFN injection. | |
| 34 | 10) Blood sample for storage (10 mL of blood separated into serum and stored frozen in 0.5-1 | .0 |
| 35 | mL aliquots) | |
| 36 | 11) Start peginterferon 180 ug SQ | |

| 1 | 12] | Repeat liver biopsy 6 hours after first dose of peginterferon. Liver biopsy cut into four |
|---|---|---|
| 2 | | sections, one (at least 1.5 cm) placed in formalin for routine light microscopy and the other $3$ |
| 3 | | (.3cm, .5cm and 1 cm) placed in RNAlater and flash frozen in liquid nitrogen 24 hours later |
| 4 | | for RNA and protein analyses and flow cytometry. |
| 5 | | |
| 6 | | |
| 7 | | |
| 8<br>9 | <u>Day1</u><br>1) | 24h after the first PegIFN injection: 50 mL of blood in heparinized green top tubes for NK. |
| 10 | -) | This is the time point where we expect the maximal response of NK cells to PegIFN based on |
| 11 | | our previous studies [35, 36] |
| 12 | 2) | Discharge from hospital |
| 13 | 2) | Discharge from hospital |
| 15 | | |
| 14 | | |
| 15 | Week 2 | <b>2,4, 8 and 12 (± 3 days):</b> Outpatient visit |
| 16 | Each o | stpatient visit will include assessment of compliance, adverse events reporting, vital signs, |
| 17 | weight | symptoms evaluation, record of concomitant medications, drug dispensing |
| 18 | 1) | Symptom questionnaire |
| 19 | 2) | Visual analogue scale |
| 20 | 3) | Fatigue questionnaire (Promise 7) (week 2 only) |
| 21 | 4) | Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, |
| 22 | | glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline |
| 23 | | Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, |
| 24 | | white blood cell count and differential, platelet count). |
| 25 | 5) | HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs measurment |
| 26 | 6) | Blood sample for storage (10 mL of blood separated into serum and plasma stored frozen in |
| 27 | | 0.5-1.0 mL aliquots) |
| 28 | 7) | 50 mL of blood in heparinized green top tubes for NK and T cell analysis. |
| 29 | 8) | Females of child bearing potential: Pregnancy test |
| 30 | 9) | TSH and quantitative HBe and HBs antigen measurement at week 12. |
| 31 | | |
| 32 | | |
| 33 | End of | Add-on Peginterferon Treatment (Week 24 ± 3 days) |
| 34 | At wee | k 24, all subjects will discontinue peginterferon alfa-2a add-on therapy (but continue the |
| 35 | NUCs a | nd undergo the following evaluation: |

| 1 | 1) | Physical examination |
|---|---|---|
| 2 | 2) | Symptom questionnaire |
| 3 | 3) | Fatigue questionnaire (Promise 7) |
| 4 | 4) | Visual analogue scale |
| 5 | 5) | Assessment of adverse events, concomitant medications and adherence |
| 6 | 6) | Blood will be drawn for Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, |
| 7 | | phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, |
| 8 | | CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC |
| 9 | | (hematocrit, hemoglobin, white blood cell count and differential, platelet count). |
| 10 | 7) | 50 mL of blood in heparinized green top tubes for NK and T cell analysis. |
| 11 | 8) | Urine tests: routine urinalysis and creatinine, phosphate and beta-2-microglobulin |
| 12 | 9) | HBV DNA viral load, HBeAg, anti-HBe, HBsAg, anti-HBs and quantitative HBe and HBs |
| 13 | | measurement |
| 14 | 10) | Blood sample for storage (10 mL of blood separated into serum and plasma stored frozen in |
| 15 | | 0.5-1.0 mL aliquots) |
| 16 | 11) | Females of child bearing potential: Pregnancy test |
| 17 | 12) | TSH |
| 10 | | |
| 1 🗙 | | |
| 18<br>19 | Doct-tr | eatment weeks 12 24 36 (+ 5 days) |
| 19 | | eatment weeks 12, 24, 36 (± 5 days) |
| 19<br>20 | 1) | Limited clinical evaluation |
| 19<br>20<br>21 | 1)<br>2) | Limited clinical evaluation Symptom questionnaire |
| 19<br>20<br>21<br>22 | 1)<br>2)<br>3) | Limited clinical evaluation Symptom questionnaire Visual analogue scale |
| 19<br>20<br>21<br>22<br>23 | 1)<br>2) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, |
| 19<br>20<br>21<br>22<br>23<br>24 | 1)<br>2)<br>3) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, |
| 19<br>20<br>21<br>22<br>23<br>24<br>25 | 1)<br>2)<br>3) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26 | 1)<br>2)<br>3)<br>4) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27 | 1)<br>2)<br>3)<br>4) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28 | 1)<br>2)<br>3)<br>4) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29 | 1)<br>2)<br>3)<br>4)<br>5)<br>6) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots) |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29<br>30 | 1)<br>2)<br>3)<br>4) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29 | 1)<br>2)<br>3)<br>4)<br>5)<br>6) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots) |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29<br>30 | 1)<br>2)<br>3)<br>4)<br>5)<br>6) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots) |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29<br>30<br>31 | 1)<br>2)<br>3)<br>4)<br>5)<br>6) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots) |
| 19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29<br>30<br>31 | 1)<br>2)<br>3)<br>4)<br>5)<br>6) | Limited clinical evaluation Symptom questionnaire Visual analogue scale Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC (hematocrit, hemoglobin, white blood cell count and differential, platelet count). HBV DNA viral load, HBeAg, anti HBe, HBsAg and anti HBs levels Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots) 50 mL of blood in heparinized green top tubes for NK and T cell analysis. |

- 1 3) Fatigue questionnaire (Promise 7) 2 4) Visual analogue scale 3 5) Routine blood panel: Chemistry 20 (sodium, chloride, potassium, bicarbonate, calcium, 4 phosphate, magnesium, glucose, blood urine nitrogen, creatinine, uric acid, ALT, AST, LDH, 5 CPK, Alkaline Phosphatase, total and direct bilirubin, albumin, total protein), CBC 6 (hematocrit, hemoglobin, white blood cell count and differential, platelet count). 7 6) Extended blood panel: alpha fetoprotein, gGT, immunoglobulins, rheumatoid factor, ANA, 8
  - SMA, lipid panel, INR, reticulocyte count, ESR.
  - 7) 50 mL of blood in heparinized green top tubes for NK and T cell analysis.
  - 8) HBV DNA viral load, HBeAg, anti HBe, HBsAg, and anti HBs levels and quantitative HBe and HBs measurement
  - 9) Blood sample for storage (10 mL of serum and 10 ml of plasma stored frozen in 0.5-1.0 mL aliquots)
  - 10) Fibroscan

16

17

9

10

11

12

Table 1: List of study related procedures

| Procedure | Screen | Pre-Rx<br>biopsy | Day 0 | Wk 2, 4, | Wk<br>12 | Week<br>24<br>End<br>of Rx | Post-<br>Rx wk<br>12, 24,<br>36 | Post-Rx<br>wk 48,<br>End of<br>Study |
|---|---|---|---|---|---|---|---|---|
| H&P/breif clinical<br>evaluation, compliance,<br>AE, concommit. drugs, | | | | | | | | |
| etc | Х | Х | Х | Х | Х | Х | Х | Х |
| Symptom questionnaire | Х | Х | Х | Х | Х | Х | Х | Х |
| Visual Analog Scale | Х | Х | Х | х | Х | Х | Х | Х |
| Promis 7 | Х | Х | Х | wk 2 | | Х | | Х |
| Chem 20 | Х | Х | Х | Х | Х | Х | Х | Х |
| CBC | Х | Х | Х | Х | Х | Х | Х | Х |
| Anti-HAV | Х | | | | | | | |
| HBsAg | Х | Х | Х | Х | Х | Х | Х | Х |
| HBsAg quantitative | | | Х | | Х | Х | | Х |
| anti-HBs | Х | | | | | | | |
| HBeAg | Х | Х | Х | Х | Х | Х | Х | Х |
| HBeAg quantitative | | | Х | | Х | Х | | Х |
| anti-HBe | Х | | | | | | | |
| anti-HBc | Х | | | | | | | |

| anti-HCV | Х | | | | | | | |
|-------------------------|-----|-------|------|-----|-----|-----|-----|-----|
| IL28B | Х | | | | | | | |
| HBV DNA | Х | Х | Х | Х | Х | Х | Х | Х |
| AFP | Х | | | | | | | Х |
| gGT | Х | | | | | | | Х |
| Immunoglobulins | Х | | | | | | | Х |
| rheumatoid factor | Х | | | | | | | Х |
| ANA | Х | | | | | | | Х |
| SMA | Х | | | | | | | Х |
| Lipid panel | Х | | | | | | | Х |
| thyroid panel | Х | | | | TSH | TSH | | |
| INR | Х | | | | | | | Х |
| reticulocyte | Х | | | | | | | Х |
| ESR | Х | | | | | | | Х |
| storage - 5mL serum and | | | Seru | | S& | | | |
| 5mL plasma | S&P | Serum | m | S&P | Р | S&P | S&P | S&P |
| Immunology - 50mL | Х | Х | Х | Х | Х | Х | | Х |
| Urine pregnancy | Х | | Х | Χ | Х | Χ | | |
| UA | Х | | | | | Χ | | |
| Urine creatinine, | | | | | | | | |
| phosphate, beta-2- | | | | | | v | | |
| microglubulin | | | Time | | | Х | | |
| Liver Biopsy | | Х | d | | | | | |
| Abdominal u/s | | Х | | | | | | |
| CXR | | Х | | | | | | |
| EKG | | Х | | | | | | |
| Fibroscan | Х | | | | | | | Х |

## **ASSESSMENT OF RESPONSE**

## **Clinical Definitions**

 a) Loss of HBeAg (HBeAg-positive patients only): loss of detectable HBeAg with or without anti-HBe seroconversion confirmed on 2 consecutive visits at least 12 weeks apart.

b) **Loss of HBsAg**: Loss of HBsAg, with or without anti HBs seroconversion confirmed on 2 consecutive visits at least 12 weeks apart.

| 1 | c) | Sustained response: virological, serological, biochemical, or combined response present at |
|---|---|---|
| 2 | Cj | |
| | | the time of last observation and at least six months after stopping therapy. |
| 3 | | |
| 4 | | |
| 5 | The primary goals of this study are centered on understanding the mechanisms, and identification of | |
| 6 | predictive factors associated with a favorable response to peginterferon therapy when added on to | |
| 7 | long-te | rm NUCs treatment, in patients with HBeAg positive and negative chronic HBV infection. |
| 8 | | |
| 9<br>L0 | Primary end-points | |
| 1 | 1) | The primary end-point for this study will be the change in level of ISG expression and NK cell |
| 12 | | responses before and after 1 <sup>st</sup> peginterferon injection in responders versus non-responders |
| 13 | | to peginterferon add-on therapy. |
| <b>L</b> 4 | 2) | Proportion of eAg positive patients showing eAg loss with or without seroconversion at end |
| 15 | | of treatment and 24 and 48 weeks off therapy. |
| 16 | 3) | Proportion of eAg positive patients showing sAg loss with or without seroconversion at end |
| 17 | , | of treatment and 24 and 48 weeks off therapy |
| 18 | 4) | Proportion of eAg negative patients showing sAg loss with or without seroconversion at at |
| 9 | , | end of treatment and 24 and 48 weeks off therapy |
| 20 | | |
| 21<br>22 | Second | lary endpoints |
| 23 | 1. | Level of qHBsAg decline at treatment week 12, at end of treatment and 24 and 48 weeks off |
| 24 | | therapy, compared to pretreatment levels in eAg positive and negative patients |
| 25 | 2. | Level of qHBeAg decline at treatment week 12, at end of treatment and 24 and 48 weeks off |
| 26 | | therapy, compared to pretreatment levels in eAg positive and negative patients |
| 27 | 3. | Correlation of qHBsAg levels at initial evaluation, week 12,24,36 and 48 with intrahepatic |
| 28 | 0. | pregenomic and cccDNA concentration before and after initiation of peginterferon in |
| 29 | | responders versus non-responders to treatment. |
| 30 | 4. | Intrahepatic pregenomic and cccDNA concentration before and after starting treatment with |
| 31 | 1. | peginterferon. |
| 32 | 5. | Epigenetic alterations in HBeAg positive and negative patients following first 1 <sup>st</sup> |
| 33 | J. | peginterferon injection compared to pretreatment levels as measured by chromatin |
| 34 | | immunoprecipitation (ChIp) assays |
| , T | | mmunopi ecipitation (cmp) assays |

1 6. Frequency and functional activity of circulating and liver infiltrating, HBV-specific T-cells, 2 measured before and during treatment in responders versus non-responders to 3 peginterferon add-on therapy. 4 5 **DOSE CHANGES** 6 7 Stopping peginterferon therapy: 8 9 Add-on peginterferon will be discontinued early for any of the following reasons: 10 a) **Toxicity**- the dose of peginterferon will be modified or discontinued according to Table 1: 11 Peg-Interferon Alfa-2a Dose Modification Guidelines (see below). 12 b) Withdrawal of informed consent (subject's decision to withdraw for any reason. 13 c) Any clinical adverse event, laboratory abnormality, or intercurrent illness, which in the 14 opinion of the investigator indicates that continued participation in the study is not in the 15 best interest of the subject. If any of the following laboratory or clinical criteria is obtained 16 for any subject, the result must be repeated/confirmed within 72 hours. If the results are 17 confirmed, the subject must discontinue treatment. Clinical criteria must have Principal 18 Investigator or Sub-Investigator assessment prior to permanent discontinuation. 19 - Evidence of confirmed hepatic decompensation (Child-Pugh Class B or C, Score > 6) 20 (discontinue all treatment); 21 Platelets  $< 25 \times 10^9 \text{ cells/L};$ 22 Hemoglobin < 8.5 g/dL 23 Absolute neutrophil count < 250 mm<sup>3</sup>/ml 24 - Severe neuropsychiatric signs and symptoms (including depression) for both new and 25 worsening events that are considered clinically significant by the investigator. 26 27 d) **Pregnancy** women of childbearing potential must contact the investigator or study staff 28 immediately if they suspect they might be pregnant (eg, missed or late menstrual period) at 29 any time during study participation. If subjects become pregnant the research staff will stop 30 peginterferon, but subjects may continue taking their antiviral oral agent at the discretion of 31 the study doctor. The investigator will discuss possible management options with the 32 subject. Subjects who do become pregnant will continue to be followed for the outcome of 33 the pregnancy. The NIH will not cover any aspects of obstetrical, child or related care.

e) Loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness.

### **Stopping NUCs therapy**

Treatment with NUCs will be stopped under the following conditions

a) HBeAg loss, with or without anti HBe seroconversion, in eAg positive patients, that is confirmed on 2 separate tests, at least 6 months apart.

b) HBsAg loss, with or without anti HBs seroconversion, that is confirmed in 2 separate tests, at least 6 months apart.

## **Peginterferon Dose Modifications**

Dose modification of peginterferon  $\alpha$ -2a should be managed according to Table 2. This table is based on recommendations from the peginterferon  $\alpha$ -2a package insert, and have been modified as necessary for this study. As Tables 2 is a guideline, investigators may modify the dose based on clinical judgment.

Table 2: Peg-Interferon Alfa-2a Dose Modification Guidelines

| Laboratory Value/Clinical | Dose Modification: | Additional Instructions: |
|---|---|---|
| Criteria: | | |
| ANC: | | |
| ≥ 0.75 × 109 cells/L | Maintain at 180 μ g | |
| ≥ 0.25 × 109 to < 0.75 × 109 | Reduce to 135 μ g | |
| cells/L | | |
| < 0.25 × 109 cells/L | All study drugs should be | Reinstitute at 90 $\mu$ g and |
| | interrupted until ANC values | monitor |
| | return to more than | ANC |
| | 1000/mm3 | |
| Platelets: | | |

| $\geq$ 50 × 10 <sup>9</sup> cells/L | Maintain at 180 μ g | |
|---|---|---|
| $\geq 25 \times 10^9 \text{ to} < 50 \times 10^9$ | Reduce to 90 µ g | |
| cells/L | | |
| < 25 × 10 <sup>9</sup> cells/L | Discontinue all study drugs if | Treatment should not be |
| | value is confirmed | reinstituted |
| ALT: | | |
| ALT > 10 × ULN | Reduce to 135 $\mu$ g or interrupt | If ALT increases are |
| | all study drugs if repeated ALT | progressive or there is |
| | results are > 10 × ULN | evidence of hepatic |
| | | decompensation therapy |
| | | should be interrupted |
| New Ocular symptom(s): | | |
| New decrease or loss of vision | Interrupt all study treatment | Complete eye examination |
| or | | must be performed. |
| other clinical significant ocular | | |
| sign or symptom | | |
| New or Worsening | Mild No change Evaluate | Evaluate weekly (with visit at |
| Neuropsychiatric Signs or | weekly by visit or phone | least every other week). |
| Symptoms (Including | until symptoms improve. | Consider psychiatric |
| Depression): | | consultation if no |
| | | mprovement. If improved and |
| | | stable for 4 weeks, may |
| | | resume normal dosing. |
| Modovato | Deduce deserts 125 | |
| Moderate | Reduce dose to 135 μ g | D. Harris |
| Severe | Discontinue all study drug | Psychiatric therapy necessary. |
| | treatment | Treatment should not be |
| | | reinstituted. |
| Creatinine Clearance (CrCl): | | |
| < 30 mL/min | Reduce to 135 μg | |
| Hemodialysis | Reduce to 135 μg | |

Source: adapted from Pegasys® package insert.

| 1 2 | STATISTICAL ANALYSIS |
|---|---|
| 3 | Power calculation |
| 5 | It is not possible to calculate power for the primary endpoints. We have calculated power for the |
| 6 | secondary endpoints of the rates of HBeAg and HBsAg loss. Response rates in patients in both groups |
| 7 | will be compared to historical controls of HBeAg positive and negative. It is assumed that if these |
| 8 | patients were followed for an additional year without peginterferon, only 10% of the HBeAg positive |
| 9 | patients would become HBeAg negative and 5% of the HBeAg negative patients would become |
| 10 | HBsAg negative. A sample size of 29 HBeAg positive and 27 HBeAg negative patients will provide the |
| 11 | study with a statistical power of $80\%$ to detect a difference of $25\%$ ( $35\%$ versus $10\%$ for HBeAg loss |
| 12 | and 30% versus 5% for HBsAg loss). The sample size was increased to 30 patients in each arm to |
| 13 | allow for withdrawals. |
| 14 | |
| 15 | Variables to be analyzed in association with a serological response will include: baseline ALT and |
| 16 | HBV DNA level, liver histology, HBV genotype, IL28B genotype, duration of NUC therapy, and ISG |
| 17 | levels. Patients with missing data or who drop out of the study will be considered as treatment |
| 18 | failures on an intention to treat basis. For comparison of means, Student's t-test will be used. All |
| 19 | reported p-values will be 2-sided. |
| 20 | |
| 21 | Demographics and Baseline Characteristics |
| 22<br>23 | The following will be summarized for treated subjects: |
| 24 | Demographics: age, race, gender, geographic region, ethnicity; |
| 25 | • Disease characteristics at baseline: HBV DNA level, HBV genotype, IL28B SNP genotype and |
| 26 | cirrhosis status, duration of NUC therapy; |
| 27 | • Physical measurements at baseline; height, weight, body mass index, hip and waist circumference; |
| 28 | • Laboratory tests at baseline; |
| 29 | |
| 30<br>31 | Analysis plan |
| 32 | To address the primary hypothesis that ISG levels are related to virological response to |
| 33 | peginterferon, the ISG analysis of the on treatment liver biopsy at 6 hours after the first dose of |
| 34 | interferon will be correlated with off-peginterferon serological outcome (HBeAg loss/seroconversion |
| 35 | and HBsAg loss). To address the hypothesis that ISG levels are related to HBsAg levels, the ISG |

analysis of the on treatment liver biopsy will be correlated with HBsAg levels at weeks 4, 12, 24.. The

| 1 2 | analyse | es will be stratified by HBV genotype and duration of NUC therapy. |
|---|---|---|
| 3 4 | Analysis methodology | |
| 5 | The analysis will be based on standard approaches to analysis of microarray data. Since the software | |
| 6 | and approaches change frequently in this field, we will provide a broad outline of the approach | |
| 7 | rather than detailed, specific steps. | |
| 8 | a) | We will perform quality control and background normalization of the gene array data. |
| 9 | b) | Expression value estimates will be obtained and quantile normalization and median scaling |
| 10 | | of the genes will be performed. |
| 11 | c) | A list of genes up- or down-regulated >2-fold with p>0.05 will be prepared using the |
| 12 | | following procedure: |
| 13 | | 1. For each patient, genes up- or down-regulated >2-fold in the second biopsy |
| 14 | | compared to the first will be identified. |
| 15 | | 2. Lists will be prepared of genes that are up- or down-regulated >2-fold for any of the |
| 16 | | subjects. |
| 17 | | 3. A paired t-test will be used to identify genes from this list that have a p value < 0.05 |
| 18 | | (Difference is not equal to zero). |
| 19 | | 4. The subset of the genes in (3) that are up- or down-regulated in >50% of patients in |
| 20 | | groups defined relapse and/or presence of cirrhosis will be identified. |
| 21 | | 5. This procedure will be repeated with $p < 0.01$ , but the primary analysis will be |
| 22 | | based on the genes selected using $p < 0.05$ . |
| 23 | d) | The false discovery rate (FDR) of the t test will be estimated. |
| 24 | A more | detailed statistical analysis plan will be developed prior to the start of data analysis. |
| 25 | | |
| 26 | | |
| 27<br>28 | | HAZARDS AND DISCOMFORTS |
| 28<br>29 | The risks and discomforts of frequent phlebotomy. | |
| 30 | To doci | ument stable levels of biochemical and serologic markers of chronic hepatitis and to monitor |

To document stable levels of biochemical and serologic markers of chronic hepatitis and to monitor the effects and toxicities of the combination of peginterferon alfa-2a and the nucleos(t)ide analogue frequent blood sampling will be required. Patients will have between 11 and 12 venipunctures during the study. Each venipuncture will be for approximately 20 to 75 cc of blood. The total amount of blood drawn during an 8 week period will not exceed 10.5 ml/Kg or 550 mls, whichever is smaller.

The risks and discomforts of HIV testing.

Patients will have blood tested for anti-HIV at entry. Mention of anti-HIV is made in the consent form which includes the exact language used in the standard consent form used for anti-HIV testing at the Clinical Center. It is important to test for HIV infection as many of the drugs used to treat hepatitis B (tenofovir, tenofovir and emtricitabine, lamivudine and entecavir) have activity against HIV and a treatment regimen using only two drugs against HIV would not be considered standard of care.

6 7

8

9

10

11

12

13

14

15

16

17

18

19

20

21

22

23

24

25

1

2

3

4

5

## The risks and discomfort of percutaneous liver biopsy.

Patients will undergo up to two liver biopsies in this protocol: one before therapy and a second six hours after the initial injection of peginterferon alfa-2a. Patients with inadequate platelet counts (<70,000/mm<sup>3</sup>) or coagulation parameters (prothrombin time > 15 seconds, INR>1.7) will undergo transjugular liver biopsy after correction of the laboratory abnormalities as a part of this protocol. Patients requiring liver biopsy will be admitted to the Clinical Center for two days for this procedure and other blood testing. The major side effects of liver biopsy are pain, bacteremia, puncture of another organ and bleeding. Local pain and discomfort at the liver biopsy site occurs in about 20% of persons undergoing percutaneous liver biopsy. This is transient (lasting one to twelve hours) and is usually mild, rarely requiring analgesics. Bacteremia occurs in 1-2% of persons undergoing liver biopsy. In the absence of bile duct obstruction, this is almost always self-limited and is rarely symptomatic. Significant bleeding after liver biopsy is the most serious side effect of this procedure. In the absence of a blood coagulation defect or hepatic malignancy, significant bleeding is rare, occurring in less than one in a thousand cases of liver biopsy. Death due to bleeding after liver biopsy has been reported in less than 1/10,000 cases. At the NIH Clinical Center, the Liver Diseases Branch has performed approximately 150 liver biopsies each year for the last 20 years. During this time, only two patients died as a complication of biopsy. One of these patients had cirrhosis and advanced hepatocellular carcinoma and the second had severe coagulation disorders. Both bled from the liver biopsy site and died after surgical attempts to stop the bleeding were unsuccessful.

2627

31

32

33

34

35

36

37

#### The risks and hazards of Peginterferon therapy

Local pain and erythema at the site of subcutaneous injection. This is usually mild and is no greater
 than the pain and irritation associated with other subcutaneous injections. Severe local reactions
 have been described but are rare

A syndrome of fever, malaise, headaches and muscle aches. These influenza- like symptoms occur typically after the first injection and decrease in severity with subsequent treatments. Fever can be as high as 40°C. The fatigue often persists or reappears with prolonged therapy with interferon and is often the dose-limiting factor in therapy. These symptoms abate with discontinuation of treatment, but may last for up to 2 weeks after the final injection of interferon. There is considerable variation in the occurrence and severity of these symptoms.

Gastrointestinal symptoms of nausea, vomiting, diarrhea and anorexia are common with high doses

1 of interferon. These are rarely severe enough to warrant discontinuation or alteration in interferon 2 therapy. 3 4 Hair loss is noted by 20-25% of patients treated with interferon for more than two months. This is 5 always temporary. 6 7 Bone marrow suppression occurs with the dose of interferon used to treat chronic hepatitis. 8 Leukopenia and granulocytopenia are the most frequent findings and a 20-50% decrease in white 9 blood cell counts is typical during therapy. This effect is always temporary and is dose related. 10 Folliculitis and sinusitis, as well as more serious infections such as dissemination of cellulitis and 11 bacterial peritonitis have occurred in patients receiving interferon. Indeed, among the more than 400 12 patients with chronic viral hepatitis treated with alpha interferon at the NIH, two died of infections 13 (spontaneous bacterial peritonitis) during therapy. Both patients had hepatitis B and end-stage liver 14 disease. Spontaneous bacterial peritonitis is a common complication of end-stage liver disease. Other 15 instances of severe and rare forms of infection have been reported in patients receiving interferon. It 16 appears that most of these severe infections are more related to the underlying condition than the 17 leukopenia induced by interferon, but interferon may increase susceptibility to infections and severe 18 outcomes. For these reasons, all patients will be cautioned, about infectious complications and 19 advised to contact their physician or the investigators if they develop fever. Thrombocytopenia also 20 occurs with interferon treatment, the platelet count falling by 13-52% of the pretreatment values. 21 Serious bleeding episodes have not been reported with interferon therapy. Finally, mild anemia with 22 a decrease in hematocrit and hemoglobin of 3-5% is also seen commonly with interferon therapy. 23 The effects of interferon on the bone marrow have been temporary and rapidly reversible with 24 discontinuation of therapy. 25 26 Significant cardiac side effects have included idiopathic and reversible heart failure. This is reversible 27 with conventional management. This occurs with a frequency of <1%. 28 29 Pulmonary disorders: Dyspnea, pulmonary infiltrates, pneumonia, bronchiolitis obliterans, 30 interstitial pneumonitis and sarcoidosis, some resulting in respiratory failure and/or patient deaths, 31 may be induced or aggravated by interferon therapy. Pulmonary complications are rare and occur 32 with a frequency of <1%. 33 34 Altered liver enzymes: Interferon can cause mild elevations in serum aminotransferases in patients 35 who do not have liver disease. In patients with chronic viral hepatitis, these possible elevations in 36 aminotransferases may be obscured by the pre-existing liver disease. Transient ALT elevations are 37 common during hepatitis B therapy with interferon. Twenty-five percent and 27% of subjects

experienced elevations of 5 to 10 x ULN and 12% and 18% had elevations of greater than 10 x ULN during treatment of HBeAg negative and HBeAg positive disease, respectively. Flares have been accompanied by elevations of total bilirubin and alkaline phosphatase and less commonly with prolongation of PT and reduced albumin levels. Eleven percent of subjects had dose modifications due to ALT flares and less than 1% of subjects were withdrawn from treatment. Of note these data refer to patients not receiving concomitant oral antiviral agents. We believe the chance of significant ALT flares (>10x ULN) would be rare in the setting of combination therapy.

Renal effects: Interferon may have minor renal toxicities. A case of interstitial nephritis during alpha interferon therapy has been reported. We have had one patient develop acute renal failure while on alpha interferon. This was only partially reversible. We have treated many patients with renal disease using alpha interferon without any adverse effects on renal function. Renal complications are rare and occur with a frequency of <1%.

CNS Effects: Confusion has been noted with very high doses of interferon (>50 mu)69. At the doses used in our trials (180 mcg per injection) the only central nervous system side effects have been mild headaches, irritability, depression and psychological changes. Many patients complain of being short-tempered and irritable while on interferon. Approximately 18% of patients develop emotional lability and depression. These side effects are closely monitored and reverse with decrease in the interferon dosage. Another 5% of patients treated with interferon in our studies developed more severe psychiatric side effects including paranoia, delusional thinking and marked anxiety. We have found this side effect largely in patients with pre-existing psychiatric or neurological problems6. These side effects reverse within one to two weeks after discontinuing interferon therapy.

<u>Seizures</u> may occur in patients receiving alpha interferon. These have been described as grand mal seizures that were self-limited and stopped once interferon was discontinued. We have reported that there is a 1-2% incidence of seizures during interferon therapy. These seizures occurred near the end of therapy and did not recur. Several patients were hospitalized for the seizures and evaluated; no abnormalities were detected on neurological examination or imaging studies, and none are currently receiving anti-epileptic medication.

Neuropsychiatric: Life-threatening or fatal neuropsychiatric reactions may manifest in all patients receiving therapy with interferon and may include suicide, suicidal ideation, homicidal ideation, relapse of drug addiction, and drug overdose. These adverse effects occur in <1% of treated subjects. These reactions may occur in patients with and without previous psychiatric illness.

myositis, hepatitis, thrombotic thrombocytopenic purpura, idiopathic thrombocytopenic purpura,
 psoriasis, rheumatoid arthritis, interstitial nephritis, thyroiditis, and systemic lupus erythematosus

O

DICE

# RISK/DISCOMFORTS IN RELATION TO BENEFIT

have been reported in patients receiving alpha interferon. These occur in less than 1% of patients.

Autoimmune phenomena: Development or exacerbation of autoimmune disorders including

**Protection against risks** 

The risks of study medication regimen administration can be generalized into 3 areas, teratogenicity, changes in hematological parameters, and non-specific side effects. To protect subjects from teratogenicity, pregnancy tests will be performed every 2 weeks for the first 2 months, then every month thereafter. Additionally, women should practice 2 forms of contraception. CBC's will be performed every 2 weeks to monitor for hematologic changes, and symptoms or side effects will be monitored at every visit, which may result in a study medication regimen dose modification. Another major risk to subjects who agree to participate in this study is the risk of undergoing 2 liver biopsies (as outlined in Risks and hazards #3). Since a major endpoint of the study is to understand how peginterferon may lead to HBeAg or HBsAg loss, the timing of the biopsies were chosen to maximize our ability to demonstrate changes in interferon stimulated genes in the liver-up to 12 weeks before and 6 hours after the first dose of peginterferon. Knowledge gained from this analysis may inform on how best to use peginterferon in patients with chronic hepatitis B and identify new approaches to induce HBeAg and HBsAg loss-highly desirable endpoints that may permit cessation of treatment.

**Potential benefits** 

For patients with chronic hepatitis B, the strategy of add-on peginterferon offers a potential benefit of loss of either HBeAg or HBsAg or both with the possibility of discontinuing all therapy and removal of the risks associated with long term nucleoside analogue use-predominantly renal toxicity and bone loss with tenofovir and cancer risk with entecavir. Thus, there is a prospect of overall clinical benefit from participation in this study.

#### **DATA AND SAFETY MONITORING**

The adequacy of data acquisition and storage of samples and the monitoring of safety in this trial will be performed by the principal investigator in collaboration with the associate investigators. Data and safety are reviewed weekly in clinical research rounds by the Liver Diseases Branch, NIDDK. These rounds are separate from regular clinical rounds and consist of review of all study patients including

1 flow sheets of major safety and efficacy measurements without knowledge of which therapy is used. 2 Monitoring of this study will also be conducted by the statistical department of NIDDK who will have 3 knowledge of the patient allocation. Reports of serious adverse events are made to the Clinical 4 Director NIDDK, and the IRB as outlined below. 5 6 ADVERSE EVENT REPORTING 7 8 **Definitions** 9 10 Protocol Deviation: Any change, divergence, or departure from the IRB approved research protocol. 11 Unanticipated Problem: Any incident, experience or outcome that meets all of the following criteria: 12 1. Unexpected (in terms of nature, severity or frequency) given (a) the research procedures 13 that are described in the protocol-related documents, such as the IRB approved research protocol 14 and informed consent document; and (b) the characteristics of the subject population being studied. 15 2. Related or possibly related to participation in the research (possibly related means there 16 is a reasonable possibility that the incident, experience or outcome may have been caused by the 17 procedures involved in the research); and 18 3. Suggests that the research places subjects or others at a greater risk of harm (including 19 physical, psychological, economic or social harm) than was previously known or recognized). 20 Expected Adverse Events become unanticipated problems when they occur at a greater frequency or 21 severity than was previously known. 22 23 Adverse events, protocol deviations, unanticipated problems (UP), Unanticipated Adverse Device 24 Effects (UADEs), serious adverse events, sponsor and serious, are defined as described in NIH HRPP 25 SOP 16 ("Reporting Requirements for Unanticipated Problems, Adverse Events and Protocol 26 Deviations."). All adverse events at least possibly related to the patient's participation in the 27 research protocol, including those observed by or reported to the research team, will be recorded. 28 Serious unanticipated problems and serious protocol deviations will be reported to the IRB and CD 29 as soon as possible but not more than 7 days after the PI first learns of the event. Not serious 30 unanticipated problems will be reported to the IRB and CD as soon as possible but not more than 14 31 days after the PI first learns of the event. 32 33 Non-serious protocol deviations will only be reported to the IRB (within 14 days after the PI first 34 learns of the event) if they represent a departure from NIH policies for the conduct of human subjects

research, adversely affect the health care of the subject(s) or compromise the interpretation or

integrity of the research. Non-serious protocol deviations that result from normal subject scheduling

35

variations or technical issues associated with sampling that do not impact the health of the subject or the interpretation of the study data will not be reported.

Adverse events that are expected as a part of treatment or procedures outlined in the protocol will not be reported unless they occur at a rate or severity greater than known to occur in patients undergoing the treatment or procedures. If AEs associated with the treatment and procedures in the study occur at a rate or severity greater than known to occur, they will be reclassified as a UP and reported as such. AEs with known relation to the natural history of chronic hepatitis B or to other pre-existing conditions will not be reported unless they occur at a rate or severity greater than known to occur in patients with hepatitis B or the subject's other pre-existing conditions. AEs that are unrelated to the research will not be reported. The PI is responsible for summarizing all reportable serious adverse events and adverse events at least possibly related at the time of Continuing Review. Deaths will be reported to the Clinical Director and IRB within 7 days after the PI first learns of the event.

## PROTOCOL MONITORING PLAN

Study procedures will be subject to audits and/or monitoring visits to ensure compliance with the protocol and applicable regulatory requirements consistent with the Liver Diseases Branch quality assurance program plan. Audit and/or monitoring visits results will be reported to the Principal Investigator for further reporting as appropriate. Study documents and pertinent hospital or clinical records will be reviewed to verify that the conduct of the study is consistent with the protocol plan.

## ENROLLMENT OF CHILDREN, WOMEN AND MINORITY INDIVIDUALS

The current protocol excludes children (age limit > 18 years) as the Liver Diseases Branch does not currently treat children. The number of children on long-term nuclos(t)ide analogue therapy would expected to be small and the requirement for two liver biopsies may be prohibitive.

Chronic HBV infection is about twice as common among men than women. We expect to include women in the proportions that occur in this disease. Thus, we expect 30% to 40% of patients to be women. The exclusion of women interested in getting pregnant or who are not able to practice adequate birth control would be the only possible bias introduced in attaining adequate representation of women in this study.

The distribution of minority individuals in our ongoing hepatitis B study (07-DK-0207) are as follows: 73% of subjects were considered minorities, 82% of whom were Asian and 14% African-American based on self-reported race and ethnicity and NIH, HHS guidelines for defining minority race. Thus, we believe minority individuals will be adequately represented in this study.

Additional Potentially Vulnerable Subject Populations

This study does not plan to accrue subjects who are prisoners nor adults who are or may be unable to provide consent. These populations are excluded as this is a more than minimal risk study due to the requirement for two liver biopsies. NIH employees are not categorically recruited, but in the event that an eligible subject presents who happens to be an NIH employee, we will follow the guidelines outlined in the inclusion of employees in NIH intramural research studies.

## RESEARCH USE, STORAGE AND DISPOSITION OF HUMAN SAMPLES AND DATA

Patients will have serum stored from selected time points during this study. These specimens will be used for repeat virological testing and special tests as needed (such as for viral levels, or measurement of serum levels of cytokines or interferon induced genes). Samples may be used to assess factors associated with response or non-response to antiviral therapy. Liver biopsy tissue may be stored if residual tissue is available after samples are taken for routine histological staining and evaluation, ISG determination and immunological testing. ISG and immunological determination will be evaluated in the Liver Diseases Branch and the routine histological evaluation by the surgical pathology services of the Clinical Center. Patient participation in this study will be kept confidential. No one other than study personnel at the clinic will be given the subject's name, address, and other personal identifying information. Some study-related forms such as the consent form will be kept in the medical record and have subject name and other personal identifying information on it. Other research forms such as study diaries and flowsheets will also contain subject name and personal identifying information. These records will be kept in locked files or computers that are password protected. Liver tissue samples will be stored in the pathology department and will have personal identifying information on it. However, other study material such as blood samples will be labeled with only an identifying number and code. Any study material that may be shared with investigators outside the NIH will not contain any personal identifying information. Only the study personnel at

the Liver Diseases Branch, Clinical Center can link your name or other personal identifiers to this code. We plan to collaborate with Dr. Gavin Cloherty, Abbott Diagnostics, to obtain the quantitative HBsAg testing, specified as a secondary aim of this study. Dr. Cloherty will receive ten to eleven 250 ul aliquots of sera from each subject for quantitative HBsAg testing. The results will be used for research and as part of a planned publication.

Research records and data as well as liver biopsy slides, biopsy reports, liver tissue and sera with the patient's name and a unique identifier will be stored indefinitely in our locked offices and freezers, the medical record department and the pathology department. These materials will be protected and tracked by standard operating procedures in the medical record and pathology departments as well as a compulsive filing system in our locked offices and freezers. There will be redundant storage of clinical information in the medical record department and our offices. Likewise, there will be redundant storage of biopsy information and materials in the pathology department and our offices. This should minimize the risk of loss or destruction of information and specimens. If that were to occur we would report it to the IRB. We do not plan to destroy this personal medical information or the liver biopsy specimens or research subject sera after completion of the study because it may be critically important for physicians (here or elsewhere) to have access them when caring for these patients in the future.

#### **RECRUITMENT PLAN**

Potentially eligible HBeAg positive and HBeAg negative subjects evaluated under protocol 91-DK-0214 and 07-DK-0207 will be informed of this trial and offered enrollment in this study. It is anticipated that the majority of subjects ( $\sim$ 85%) will be recruited from within the Liver Diseases Branch Outpatient Clinic. For the remaining subjects, we will plan to send a recruitment letter to area Internists and Gastroenterologists to refer suitable candidates for the trial. Finally, we will advertise through the NIH patient recruitment office. All recruitment material will be submitted to the IRB review prior to dissemination.

#### PRIVACY AND CONFIDENTIALITY

Potentially eligible subjects will be identified through their enrolment in 91-DK-0214 and 07-DK-0207 and will be informed of this study at the time of a scheduled visit or by phone to notify them of their potential eligibility. Subjects will discuss protocol eligibility with the principal investigator or an associate investigator, and associate investigators will continue to be involved in research activities throughout subjects' participation in this study. Information collected about subjects will be obtained through routine clinical interactions including documentation in the subjects' medical

charts and through questionnaire completion, patient diaries and telephone calls. We will verbally verify with subjects their partner's compliance with subject reported reproductive contraception use, but this information will not be documented in the subjects' medical charts as these individuals are not considered subjects under this study. The information collected from subjects is primarily required to manage the subjects' clinical care under the current study. Data collected for research only is the minimal information required to complete analysis for primary and secondary aims.

#### CONSENT PROCESS

Potential study subjects will be informed of study rationale, design, participation burden, risks, benefits and side effects of therapy during routine LDB clinic visits and will have an opportunity to ask questions about the proposed study. They will be provided a copy of the study consent form to take home and review in more detail. Consent will be obtained by the Principal Investigator, or an Associate Investigator following the subject's review of the provided consent documentation during a subsequent clinic visit. If a subject indicates a desire to participate in the research study, he/she will have all screening laboratories, radiologic imaging and if necessary, liver biopsy, performed through this protocol. The initial liver and second liver biopsy for participation in this study will be for research purposes. Patients who refuse either liver biopsy will be excluded from further participation in the study, since one of the primary endpoints of the trial is based on analysis of change in ISG levels comparing the second to the first liver biopsy. Potential study subjects who meet study inclusion and exclusion criteria will sign the consent form to participate in this study during a scheduled LDB clinic visit prior to screening.

We do not plan to enroll non-English speaking subjects; however they are not excluded from participation either. Should a non-English speaking subject be enrolled, IRB approval will be obtained to use the short form process in the absence of a fully translated consent document. Requests for IRB approval will be obtained prior to implementing the short form consent process. The short form consent process will be incompliance with SOP 12.9.1 and 45 CFR 46.117(b)(2).

 **COMPENSATION** 

- 1 Patients enrolled in this trial will not be offered compensation since they will be receiving study
- 2 medications and all required monitoring at no personal cost. In addition patients stand to derive
- 3 clinical benefit from participation in the study.

# 5 REFERENCES

- Lok, A.S. and B.J. McMahon, *Chronic hepatitis B: update 2009.* Hepatology,
   2009. 50(3): p. 661-2.
- 9 2. Goldstein, S.T., et al., *A mathematical model to estimate global hepatitis B*10 *disease burden and vaccination impact.* Int J Epidemiol, 2005. **34**(6): p. 132911 39.
- 12 3. Chen, C.J., et al., *Risk of hepatocellular carcinoma across a biological gradient* of serum hepatitis *B virus DNA level.* JAMA, 2006. **295**(1): p. 65-73.
- 4. McMahon, B.J., *Natural history of chronic hepatitis B.* Clin Liver Dis, 2010.
  14 (3): p. 381-96.
- 5. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol, 2012. 57(1): p. 167-85.
- 18 6. Liaw, Y.F., et al., *Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2005 update.* Liver Int, 2005. **25**(3): p. 472-89.
- 7. Chang, T.T., et al., Long-term entecavir therapy results in the reversal of fibrosis/cirrhosis and continued histological improvement in patients with chronic hepatitis B. Hepatology, 2010. **52**(3): p. 886-93.
- 8. Marcellin, P., et al., Regression of cirrhosis during treatment with tenofovir
   disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up
   study. Lancet, 2013. 381(9865): p. 468-75.
- Hadziyannis, S.J., et al., Efficacy of long-term lamivudine monotherapy in patients with hepatitis B e antigen-negative chronic hepatitis B. Hepatology,
   2000. 32(4 Pt 1): p. 847-51.
- Hadziyannis, S.J., et al., *Long-term therapy with adefovir dipivoxil for HBeAg*negative chronic hepatitis B. N Engl J Med, 2005. **352**(26): p. 2673-81.
- Shouval, D., et al., Relapse of hepatitis B in HBeAg-negative chronic hepatitis B patients who discontinued successful entecavir treatment: the case for continuous antiviral therapy. J Hepatol, 2009. 50(2): p. 289-95.
- Chang, T.T., et al., Entecavir treatment for up to 5 years in patients with
   hepatitis B e antigen-positive chronic hepatitis B. Hepatology, 2010. 51(2): p.
   422-30.
- 37 13. Marcellin, P., et al., Long-term efficacy and safety of adefovir dipivoxil for the treatment of hepatitis B e antigen-positive chronic hepatitis B. Hepatology, 2008. **48**(3): p. 750-8.
- 40 14. Liaw, Y.F., et al., 2-Year GLOBE trial results: telbivudine Is superior to
   41 lamivudine in patients with chronic hepatitis B. Gastroenterology, 2009.
   42 136(2): p. 486-95.

- 1 15. Marcellin, P., et al., *Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B.* N Engl J Med, 2008. **359**(23): p. 2442-55.
- Fung, J., et al., Extrahepatic effects of nucleoside and nucleotide analogues in chronic hepatitis B treatment. J Gastroenterol Hepatol, 2014. 29(3): p. 428-34.
- Lu, J., et al., *Direct economic burden of hepatitis B virus related diseases:* evidence from Shandong, China. BMC Health Serv Res, 2013. **13**: p. 37.
- 8 18. Rifkin, B.S. and M.A. Perazella, *Tenofovir-associated nephrotoxicity: Fanconi syndrome and renal failure.* Am J Med, 2004. **117**(4): p. 282-4.
- 10 19. Toy, M., et al., *The cost-effectiveness of treating chronic hepatitis B patients in a median endemic and middle income country.* Eur J Health Econ, 2012. **13**(5): p. 663-76.
- Tsai, N., et al., *Cost-effectiveness of entecavir versus adefovir for the treatment*of chronic hepatitis B in patients with decompensated cirrhosis from a thirdparty US payer perspective. Clinicoecon Outcomes Res., 2012. 4: p. 227-35.
- Lok, A.S., et al., Efficacy of entecavir with or without tenofovir disoproxil fumarate for nucleos(t)ide-naive patients with chronic hepatitis B.
   Gastroenterology, 2012. 143(3): p. 619-28 e1.
- Janssen, H.L., et al., *Pegylated interferon alfa-2b alone or in combination with lamivudine for HBeAg-positive chronic hepatitis B: a randomised trial.* Lancet, 2005. **365**(9454): p. 123-9.
- 22 23. Lau, G.K., et al., *Peginterferon Alfa-2a, lamivudine, and the combination for HBeAg-positive chronic hepatitis B.* N Engl J Med, 2005. **352**(26): p. 2682-95.
- 24 24. Marcellin, P., et al., *Peginterferon alfa-2a alone, lamivudine alone, and the two in combination in patients with HBeAg-negative chronic hepatitis B.* N Engl J Med, 2004. **351**(12): p. 1206-17.
- 25. Piccolo, P., et al., A randomized controlled trial of pegylated interferon-alpha2a
   28 plus adefovir dipivoxil for hepatitis B e antigen-negative chronic hepatitis B.
   29 Antivir Ther, 2009. 14(8): p. 1165-74.
- 30 26. Bonino, F., et al., *Predicting response to peginterferon alpha-2a, lamivudine* 31 and the two combined for HBeAg-negative chronic hepatitis B. Gut, 2007. 32 **56**(5): p. 699-705.
- 33 27. Tseng, T.C., et al., Effect of host and viral factors on hepatitis B e antigen-34 positive chronic hepatitis B patients receiving pegylated interferon-alpha-2a 35 therapy. Antivir Ther, 2011. **16**(5): p. 629-37.
- 36 28. al, S.M.J.X.Q.Z.N.P.e., Adding peginterferon alfa-2a to entecavir increases HBsAg
   37 decline and HBeAg clearance first results from a global randomized trial
   38 (ARES study). Hepatology, 2012. 56(S1): p. 199A.
- 39 29. Ouzan, D., et al., Add-on peg-interferon leads to loss of HBsAg in patients with 40 HBeAg-negative chronic hepatitis and HBV DNA fully suppressed by long-term 41 nucleotide analogs. J Clin Virol, 2013. **58**(4): p. 713-7.
- 42 30. Sadler, A.J. and B.R. Williams, *Interferon-inducible antiviral effectors.* Nat Rev Immunol, 2008. **8**(7): p. 559-68.
- Li, J., et al., Inhibition of hepatitis B virus replication by MyD88 involves
   accelerated degradation of pregenomic RNA and nuclear retention of pre-S/S
   RNAs. J Virol, 2010. 84(13): p. 6387-99.

- Wieland, S.F., L.G. Guidotti, and F.V. Chisari, *Intrahepatic induction of alpha/beta interferon eliminates viral RNA-containing capsids in hepatitis B virus transgenic mice.* J Virol, 2000. **74**(9): p. 4165-73.
- 4 33. Xu, C., et al., *Interferons accelerate decay of replication-competent nucleocapsids of hepatitis B virus.* J Virol, 2010. **84**(18): p. 9332-40.
- Belloni, L., et al., *IFN-alpha inhibits HBV transcription and replication in cell* culture and in humanized mice by targeting the epigenetic regulation of the nuclear cccDNA minichromosome. J Clin Invest, 2012. **122**(2): p. 529-37.
- 9 35. Ahlenstiel, G., et al., Early changes in natural killer cell function indicate virologic response to interferon therapy for hepatitis C. Gastroenterology, 2011. **141**(4): p. 1231-9, 1239 e1-2.
- 12 36. Edlich, B., et al., Early changes in interferon signaling define natural killer cell 13 response and refractoriness to interferon-based therapy of hepatitis C patients. 14 Hepatology, 2012. **55**(1): p. 39-48.
- 15 37. Rehermann, B., *Pathogenesis of chronic viral hepatitis: differential roles of T cells and NK cells.* Nat Med, 2013. **19**(7): p. 859-68.
- 17 38. Lanford, R.E., et al., Genomic response to interferon-alpha in chimpanzees:
  18 implications of rapid downregulation for hepatitis C kinetics. Hepatology,
  19 2006. **43**(5): p. 961-72.
1 Appendix 1. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | | | | |
| HIV POSITIVE | 8.5 to 10.0 g/dL | 7.5 to < 8.5 g/dL | 6.5 to < 7.5 g/dL | < 6.5 g/dL |
| Adult and Pediatric | 85 to 100 g/L | 75 to < 85 g/L | 65 to < 75 g/L | < 65 g/L |
| ≥ 57 Days | | | | |
| HIV NEGATIVE | 10.0 to 10.9 g/dL | 9.0 to < 10.0 g/dL | 7.0 to < 9.0 g/dL | < 7.0 g/dL |
| Adult and Pediatric | 100 to 109 g/L | 90 to < 100 g/L | 70 to < 90 g/L | < 70 g/L |
| ≥ 57 Days | OR | o.p. | o.p. | |
| | UK | OR | OR | |
| | Any decrease | Any decrease | Any decrease | |
| | from Baseline | from Baseline | from Baseline | |
| | | nom basemie | nom basenne | |
| | 2.5 to < 3.5 g/dL | 3.5 to < 4.5 g/dL | ≥ 4.5 g/dL | |
| | | , | <i>,</i> | |
| | 25 to < 35 g/L | 35 to < 45 g/L | ≥ 45 g/L | |
| Infant, 36-56 Days | 8.5 to 9.4 g/dL | 7.0 to < 8.5 g/dL | 6.0 to < 7.0 g/dL | < 6.0 g/dL |
| (HIV POSITIVE OR | | | | |
| NEGATIVE) | 85 to 94 g/L | 70 to < 85 g/L | 60 to < 70 g/L | < 60 g/L |
| Infant, 22-35 Days | 9.5 to 10.5 g/dL | 8.0 to < 9.5 g/dL | 7.0 to < 8.0 g/dL | < 7.0 g/dL |
| (HIV POSITIVE OR | | | | |
| NEGATIVE) | 95 to 105 g/L | 80 to < 95 g/L | 70 to < 80 g/L | < 70 g/L |
| Infant, 1–21 Days | 12.0 to 13.0 g/dL | 10.0 to | 9.0 to < 10.0 g/dL | < 9.0 g/dL |
| (HIV positive or | | < 12.0 g/dL | | |
| negative) | 120 to 130 g/L | | 90 to < 100 g/L | < 90 g/L |
| | | 100 to < 120 g/L | | |
| Absolute | | | | |
| Neutrophil Count | 1000 to 1300/m | 750 to < | 500 to < | < 500/mm3 |
| (ANC) | m3 | 1000/mm3 | 750/mm3 | |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| | 1.00 to 1.30 GI/L | 0.75 to < 1.00 | 0.50 to < 0.75 | < 0.50 GI/L |
| Adult and Pediatric, | | GI/L | GI/L | |
| > 7 Days | | | | |
| Infant, 2 – ≤ 7 Days | 1250 to | 1000 to < | 750 to < | < 750/mm3 |
| | 1500/mm3 | 1250/mm3 | 1000/mm3 | |
| | | | | < 0.75 GI/L |
| | 1.25 to 1.50 GI/L | 1.00 to < 1.25 | 0.75 to < 1.00 | |
| | | GI/L | GI/L | |
| Infant, 1 Day | 4000 to | 3000 to < | 1500 to < | < 1500/mm3 |
| | 5000/mm3 | 4000/mm3 | 3000/mm3 | |
| | | | | < 1.50 GI/L |
| | 4.00 to 5.00 GI/L | 3.00 to < 4.00 | 1.50 to < 3.00 | |
| | | GI/L | GI/L | |
| Absolute CD4+ | | | | |
| Count | | | | |
| HIV NEGATIVE | | | | |
| ONLY | 300 to 400/mm3 | 200 to < 300/mm | 100 to < 200/mm | <100/mm3 |
| | | 3 | 3 | |
| Adult and Pediatric | 300 to 400/μL | | | < 100/μL |
| > 13 Years | | 200 to < 300/μL | 100 to < 200/μL | |
| Absolute | | | | |
| Lymphocyte Count | | | | |
| HIV NEGATIVE | | | | |
| ONLY | 600 to 650/mm3 | 500 to < | 350 to < | <350/mm3 |
| | | 600/mm3 | 500/mm3 | |
| Adult and Pediatric | 0.60 to 0.65 GI/L | | | < 0.35 GI/L |
| > 13 Years | | 0.50 to < 0.60 | 0.35 to < 0.50 | |
| | | GI/L | GI/L | |
| Platelets | 100,000 to | 50,000 to | 25,000 to | < 25,000/mm |
| | < 125,000/mm3 | < 100,000/mm3 | < 50,000/mm3 | 3 |
| | , | , ,,, | | |
| | 100 to < 125 GI/L | 50 to < 100 GI/L | 25 to < 50 GI/L | < 25 GI/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| WBCs | 2000/mm3 to | 1,500 to | 1000 to | < 1000/mm3 |
| | 2500/mm3 | < 2,000/mm3 | < 1,500/mm3 | |
| | 2.00 GI/L to | 1.50 to | 1.00 to | < 1.00 GI/L |
| | 2.50 GI/L | < 2.00 GI/L | < 1.50 GI/L | |
| Hypofibrinogenemi | 100 to 200 mg/dL | 75 to | 50 to < 75 mg/dL | < 50 mg/dL |
| a | | < 100 mg/dL | | |
| | 1.00 to 2.00 g/L | 0.75 to < 1.00 g/L | 0.50 to < 0.75 g/L | < 0.50 g/L |
| Hyperfibrinogenem | > ULN to | > 600 mg/dL | _ | _ |
| ia | 600 mg/dL | | | |
| | > ULN to 6.0 g/L | > 6.0 g/L | _ | _ |
| Fibrin Split Product | 20 to 40 μg/mL | > 40 to 50 μg/mL | > 50 to 60 μg/mL | > 60 μg/mL |
| | 20 to 40 mg/L | > 40 to 50 mg/L | > 50 to 60 mg/L | > 60 mg/L |
| Prothrombin Time | > 1.00 to 1.25 × | > 1.25 to 1.50 × | > 1.50 to 3.00 × | > 3.00 × ULN |
| (PT) | ULN | ULN | ULN | |
| International | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Normalized Ratio of | | | | |
| prothrombin time | | | | |
| (INR) | | | | |
| Activated Partial | | | | |
| Thromboplastin | > 1.00 to 1.66 × | > 1.66 to 2.33 × | > 2.33 to 3.00 × | > 3.00 × ULN |
| Time (APTT) | ULN | ULN | ULN | |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln< td=""><td>125 to</td><td>121 to</td><td>&lt; 121 mEq/L</td></lln<> | 125 to | 121 to | < 121 mEq/L |
| | mEq/L | < 130 mEq/L | < 125 mEq/L | |
| | 130 to <lln< td=""><td>125 to</td><td>121 to</td><td>&lt; 121 mmol/L</td></lln<> | 125 to | 121 to | < 121 mmol/L |
| | mmol/L | < 130 mmol/L | < 125 mmol/L | |
| Hypernatremia | 146 to 150 | > 150 to 154 | > 154 to 159 | > 159 mEq/L |
| | mEq/L | mEq/L | mEq/L | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| | 146 to 150 | > 150 to 154 | > 154 to 159 | > 159 mmol/L |
| | mmol/L | mmol/L | mmol/L | |
| Hypokalemia | 3.0 to 3.4 mEq/L | 2.5 to | 2.0 to | < 2.0 mEq/L |
| | | < 3.0 mEq/L | < 2.5 mEq/L | |
| | 3.0 to 3.4 | 2.5 to | 2.0 to | < 2.0 mmol/L |
| | mmol/L | < 3.0 mmol/L | < 2.5 mmol/L | |
| Hyperkalemia | 5.6 to 6.0 mEq/L | > 6.0 to | > 6.5 to | > 7.0 mEq/L |
| | | 6.5 mEq/L | 7.0 mEq/L | |
| | 5.6 to 6.0 | > 6.0 to | > 6.5 to | > 7.0 mmol/L |
| | mmol/L | 6.5 mmol/L | 7.0 mmol/L | |
| Hypoglycemia | | | | |
| Adult and Pediatric | 55 to 64 mg/dL | 40 to | 30 to | < 30 mg/dL |
| | | < 55 mg/dL | < 40 mg/dL | |
| ≥ 1 Month | 3.03 to | 2.20 to | 1.64 to | < 1.64 mmol/L |
| | 3.58 mmol/L | < 3.03 mmol/L | < 2.20 mmol/L | |
| Infant, < 1 Month | 50 to 54 mg/dL | 40 to | 30 to | < 30 mg/dL |
| | | < 50 mg/dL | < 40 mg/dL | |
| | 2.8 to | | | < 1.7 mmol/L |
| | 3.0 mmol/L | 2.2 to | 1.7 to | |
| | | < 2.8 mmol/L | < 2.2 mmol/L | |
| Hyperglycemia, | 116 to | > 160 to | > 250 to | > 500 mg/dL |
| Nonfasting | 160 mg/dL | 250 mg/dL | 500 mg/dL | |
| | 6.42 to | > 8.91 to | > 13.90 to | > 27.79 |
| | 8.91 mmol/L | 13.90 mmol/L | 27.79 mmol/L | mmol/L |
| Hyperglycemia, | 110 to 125 | >125 to 250 | >250 to 500 | >500 mg/dL |
| Fasting | mg/dL | mg/dL | mg/dL | |
| | | | | >27.79 |
| | 6.08 to 6.96 | >6.96 to 13.90 | >13.90 to 27.79 | mmol/L |
| | mmol/L | mmol/L | mmol/L | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia | | | | |
| (corrected for | 7.8 to 8.4 | 7.0 to < 7.8 | 6.1 to | < 6.1 mg/dL |
| albumin if | mg/dL | mg/dL | < 7.0 mg/dL | |
| appropriate*) | 1.94 to 2.10 | 1.74 to < 1.94 | 1.51 to < 1.74 | < 1.51 mmol/L |
| | mmol/L | mmol/L | mmol/L | , |
| Adult and Pediatric | , | , | , | |
| ≥ 7 Days | | | | |
| Infant, < 7 Days | 6.5 to 7.5 mg/dL | 6.0 to < 6.5 | 5.5 to < 6.0 | < 5.5 mg/dL |
| | | mg/dL | mg/dL | |
| | 1.61 to 1.88 | | | < 1.36 mmol/L |
| | mmol/L | 1.49 to < 1.61 | 1.36 to < 1.49 | |
| | | mmol/L | mmol/L | |
| Hypercalcemia | | | | |
| (corrected for | | | | |
| albumin if | >ULN to 11.5 | > 11.5 to 12.5 | > 12.5 to 13.5 | > 13.5 mg/dL |
| appropriate*) Adult | mg/dL | mg/dL | mg/dL | |
| and Pediatric ≥ | >ULN to 2.88 | > 2.88 to 3.13 | > 3.13 to 3.38 | > 3.38 mmol/L |
| 7 Days | mmol/L | mmol/L | mmol/L | |
| Infant, < 7 Days | 11.5 to 12.4 | > 12.4 to 12.9 | > 12.9 to 13.5 | > 13.5 mg/dL |
| | mg/dL | mg/dL | mg/dL | |
| | | | | > 3.38 mmol/L |
| | 2.86 to 3.10 | > 3.10 to 3.23 | > 3.23 to 3.38 | |
| | mmol/L | mmol/L | mmol/L | |
| Hypocalcemia | 3.0 mg/dL to < | 2.5 to < 3.0 | 2.0 to < 2.5 | < 2.0 mg/dL |
| (ionized) | LLN | mg/dL | mg/dL | |
| | 0.74 mmol/L to | 0.62 to < 0.74 | 0.49 to < 0.62 | < 0.49 mmol/L |
| | < LLN | mmol/L | mmol/L | |
| Hypercalcemia | > ULN to 6.0 | > 6.0 to 6.5 | > 6.5 to 7.0 | > 7.0 mg/dL |
| (ionized) | mg/dL | mg/dL | mg/dL | |
| | > ULN to 1.50 | > 1.50 to 1.63 | > 1.63 to 1.75 | > 1.75 mmol/L |
| | mmol/L | mmol/L | mmol/L | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypomagnesemia | 1.40 to <lln< td=""><td>1.04 to &lt; 1.40</td><td>0.67 to &lt; 1.04</td><td>&lt; 0.67 mg/dL</td></lln<> | 1.04 to < 1.40 | 0.67 to < 1.04 | < 0.67 mg/dL |
| | mg/dL | mg/dL | mg/dL | |
| | | | | < 0.6 mEq/L |
| | 1.2 to <lln< td=""><td>0.9 to &lt; 1.2</td><td>0.6 to &lt; 0.9</td><td></td></lln<> | 0.9 to < 1.2 | 0.6 to < 0.9 | |
| | mEq/L | mEq/L | mEq/L | |
| | 0.58 to <lln< td=""><td>0.43 to &lt; 0.58</td><td>0.28 to &lt; 0.43</td><td>&lt; 0.28 mmol/L</td></lln<> | 0.43 to < 0.58 | 0.28 to < 0.43 | < 0.28 mmol/L |
| | mmol/L | mmol/L | mmol/L | |
| Hypophosphatemia | | | | |
| Adult and Pediatric | 2.0 to < LLN | 1.5 to < 2.0 | 1.0 to < 1.5 | < 1.0 mg/dL |
| | mg/dL | mg/dL | mg/dL | |
| > 14 Years | 0.63 to < LLN | 0.47 to < 0.63 | 0.31 to < 0.47 | < 0.31 mmol/L |
| | mmol/L | mmol/L | mmol/L | |
| Pediatric 1 Year–14 | 3.0 to 3.5 mg/dL | 2.5 to < 3.0 | 1.5 to < 2.5 | < 1.5 mg/dL |
| Years | | mg/dL | mg/dL | |
| | 0.96 to 1.14 | | | < 0.47 mmol/L |
| | mmol/L | 0.80 to | 0.47 to < 0.80 | |
| | | < 0.96 mmol/L | mmol/L | |
| Pediatric < 1 Year | 3.5 to 4.5 mg/dL | 2.5 to | 1.5 to < 2.5 | < 1.5 mg/dL |
| | | < 3.5 mg/dL | mg/dL | |
| | 1.12 to 1.46 | | | < 0.47 mmol/L |
| | mmol/L | 0.80 to | 0.47 to < 0.80 | |
| | | < 1.12 mmol/L | mmol/L | |
| Hyperbilirubinemia | | | | |
| Adult and Pediatric | > 1.0 to 1.5 × | > 1.5 to 2.5 × | > 2.5 to 5.0 × | > 5.0 × ULN |
| > 14 Days | ULN | ULN | ULN | |
| Infant, ≤ 14 Days | NUCs | 20.0 to 25.0 | > 25.0 to 30.0 | > 30.0 mg/dL |
| (non-hemolytic) | | mg/dL | mg/dL | |
| | | | | > 513 µmol/L |
| | | 342 to 428 | > 428 to 513 | |
| | | μmol/L | μmol/L | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infant, ≤ 14 Days | NUCs | NUCs | 20.0 to 25.0 | > 25.0 mg/dL |
| (hemolytic) | | | mg/dL | |
| | | | | > 428 µmol/L |
| | | | 342 to 428 | |
| | | | μmol/L | |
| Blood Urea Nitrogen | 1.25 to 2.50 × | > 2.50 to 5.00 × | > 5.00 to 10.00 × | > 10.00 × ULN |
| | ULN | ULN | ULN | |
| Hyperuricemia | >ULN to 10.0 | > 10.0 to 12.0 | > 12.0 to 15.0 | > 15.0 mg/dL |
| | mg/dL | mg/dL | mg/dL | |
| | >ULN to 597 | > 597 to 716 | > 716 to 895 | > 895 µmol/L |
| | μmol/L | μmol/L | μmol/L | |
| Hypouricemia | 1.5 mg/dL to < | 1.0 to < 1.5 | 0.5 to < 1.0 | < 0.5 mg/dL |
| | LLN | mg/dL | mg/dL | |
| | 87 μmol/L to < | 57 to < 87 | 27 to < 57 | < 27 μmol/L |
| | LLN | μmol/L | μmol/L | |
| Creatinine | > 1.50 to 2.00 | > 2.00 to 3.00 | > 3.00 to 6.00 | > 6.00 mg/dL |
| | mg/dL | mg/dL | mg/dL | |
| | > 133 to 177 | > 177 to 265 | > 265 to 530 | > 530 µmol/L |
| | μmol/L | μmol/L | μmol/L | |
| Bicarbonate | 16.0 mEq/L to | 11.0 to < 16.0 | 8.0 to < 11.0 | < 8.0 mEq/L |
| | < LLN | mEq/L | mEq/L | |
| | 16.0 mmol/L to | 11.0 to < 16.0 | 8.0 to < 11.0 | < 8.0 mmol/L |
| | < LLN | mmol/L | mmol/L | |
| Triglycerides | NUCs | 500 to 750 | > 750 to 1200 | > 1200 mg/dL |
| | | mg/dL | mg/dL | |
| (Fasting) | | 5.64-8.47 | > 8.47-13.55 | > 13.55 |
| | | mmol/L | mmol/L | mmol/L |
| LDL | 130 to 160 | >160 to 190 | > 190 mg/dL | NUCs |
| | mg/dL | mg/dL | | |
| (Fasting) | 3.35 to 4.15 | >4.15 to 4.92 | >4.92 mmol/L | |
| | mmol/L | mmol/L | | |
| Pediatric >2 to <18 | 110 to 130 | >130 to 190 | > 190 mg/dL | NUCs |
| years | mg/dL | mg/dL | | |

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × | > 2.50 to 5.00 × | > 5.00 to 10.00 × | > 10.00 × ULN |
| | ULN | ULN | ULN | |
| ALT (SGPT) | 1.25 to 2.50 × | > 2.50 to 5.00 × | > 5.00 to 10.00 × | > 10.00 × ULN |
| | ULN | ULN | ULN | |
| GGT | 1.25 to 2.50 × | > 2.50 to 5.00 × | > 5.00 to 10.00 × | > 10.00 × ULN |
| | ULN | ULN | ULN | |
| Alkaline | 1.25 to 2.50 × | > 2.50 to 5.00 × | > 5.00 to 10.00 × | > 10.00 × ULN |
| Phosphatase | ULN | ULN | ULN | |
| Total Amylase | > 1.0 to 1.5 × | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × | > 5.0 × ULN |
| | ULN | | ULN | |
| Pancreatic | > 1.0 to 1.5 × | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × | > 5.0 × ULN |
| Amylase | ULN | | ULN | |
| Lipase | > 1.0 to 1.5 × | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × | > 5.0 × ULN |
| | ULN | | ULN | |

Calcium should be corrected for albumin if albumin is < 4.0 g/dL

| ENZYMES | | | | |
|---------|-----------------|-------------------|------------|---------|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Albumin | 3.0 g/dL to < | 2.0 to < 3.0 g/dL | < 2.0 g/dL | NUCs |
| | LLN | | | |
| | | 20 to < 30 g/L | < 20 g/L | |
| | 30 g/L to < LLN | | | |

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hematuria | 1+ | 2+ | 3-4+ | NUCs |
| (Dipstick) | | | | |
| Hematuria | | | | |
| (Quantitative) | | | | |
| See Note below | | | | |
| | >ULN - | > 10-75 RBC/HPF | > 75 RBC/HPF | NUCs |
| | 10 RBC/HPF | | | |
| Females | | | | |
| | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NUCs |
| Males | | | | |
| Proteinuria | 1+ | 2-3+ | 4+ | NUCs |
| (Dipstick) | | | | |
| Proteinuria, 24 | | | | |
| Hour Collection | | | | |
| Adult and | 200 to 999 | >999 to 1999 | >1999 to 3500 | > 3500 mg/24 |
| Pediatric | mg/24 h | mg/24 h | mg/24 h | h |
| ≥ 10 Years | | | | |
| Pediatric > 3 Mo to | 201 to 499 | >499 to 799 | >799 to 1000 | > 1000 mg/ |
| < 10 Years | mg/m2/24 h | mg/m2/24 h | mg/m2/24 h | m2/24 h |
| Glycosuria | 1+ | 2-3+ | 4+ | NUCs |
| (Dipstick) | | | | |

Notes:

<sup>3</sup> Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory,

<sup>4</sup> however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.

With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and
 ULN should be assigned Grade 0.

If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| 4 |
|---|
| 5 |

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia | Asymptomatic | Asymptomatic | Symptomatic, | Life-threatening |
| (general) | AND No | AND Non- | non-life- | arrhythmia OR |
| | intervention | urgent medical | threatening | Urgent |
| (By ECG or physical | indicated | intervention | AND Non- | intervention |
| exam) | | indicated | urgent medical | indicated |
| | | | intervention | |
| | | | indicated | |
| Cardiac- | NUCs | NUCs | Symptomatic | Unstable angina |
| ischemia/Infarction | | | ischemia | OR Acute |
| | | | (stable angina) | myocardial |
| | | | OR Testing | infarction |
| | | | consistent with | |
| | | | ischemia | |
| Hemorrhage | NUCs | Symptomatic | Symptomatic | Life-threatening |
| (significant acute | | AND No | AND | hypotension OR |
| blood loss) | | transfusion | Transfusion of | Transfusion of |
| | | indicated | ≤ 2 units | > 2 units packed |
| | | | packed RBCs | RBCs indicated |
| | | | (for children | (for children |
| | | | ≤ 10 cc/kg) | ≤ 10 cc/kg) |
| | | | indicated | indicated |
| Hypertension (with | 140-159 mmHg | > 159-179 | > 179 mmHg | Life-threatening |
| repeat testing at same | systolic | mmHg systolic | systolic | consequences |
| visit) | OR | OR | OR | (eg, malignant |
| | 90-99 mmHg | > 99-109 | > 109 mmHg | hypertension) |
| | diastolic | mmHg diastolic | diastolic | OR |
| | | | | Hospitalization |
| | | | | (other than ER |
| | | | | visit) indicated |

| CARDIOVASCULAR | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pediatric ≤ 17 Years | NUCs | 91st-94th | ≥ 95th | Life-threatening |
| (with repeat testing at | | percentile | percentile | consequences |
| same visit) | | adjusted for | adjusted for | (eg, malignant |
| | | age, height, and | age, height, and | hypertension) |
| | | gender (systolic | gender (systolic | OR |
| | | and/or | and/or | Hospitalization |
| | | diastolic) | diastolic) | indicated (other |
| | | | | than emergency |
| | | | | room visit) |
| Hypotension | NUCs | Symptomatic, | Symptomatic, | Shock requiring |
| | | corrected with | IV fluids | use of |
| | | oral fluid | indicated | vasopressors or |
| | | replacement | | mechanical |
| | | | | assistance to |
| | | | | maintain blood |
| | | | | pressure |
| Pericardial Effusion | Asymptomatic, | Asymptomatic, | Effusion with | Life-threatening |
| | small effusion | moderate or | non-life- | consequences |
| | requiring no | larger effusion | threatening | (eg, tamponade) |
| | intervention | requiring no | physiologic | OR Urgent |
| | | intervention | consequences | intervention |
| | | | OR Effusion | indicated |
| | | | with nonurgent | |
| | | | intervention | |
| | | | indicated | |
| Prolonged PR Interval | PR interval | PR interval | Type II 2nd | Complete AV |
| | 0.21 to 0.25 sec | > 0.25 sec | degree AV | block |
| | | | block OR | |
| | | | Ventricular | |
| | | | pause > 3.0 sec | |

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pediatric ≤ 16 Years | 1st degree AV | Type I 2nd | Type II 2nd | Complete AV |
| | block | degree AV block | degree AV | block |
| | (PR > normal | | block | |
| | for age and | | | |
| | rate) | | | |
| Prolonged QTc | Asymptomatic, | Asymptomatic, | Asymptomatic, | Life-threatening |
| | QTc interval | QTc interval | QTc interval | consequences, |
| | 0.45 to 0.47 sec | 0.48 to 0.49 sec | ≥ 0.50 sec OR | eg, Torsade de |
| | OR Increase | OR Increase in | Increase in | pointes or other |
| | interval < 0.03 | interval 0.03 to | interval | associated |
| | sec above | 0.05 sec above | ≥ 0.06 sec | serious |
| | baseline | baseline | above baseline | ventricular |
| | | | | dysrhythmia |
| Pediatric≤16 Years | Asymptomatic, | Asymptomatic, | Asymptomatic, | Life-threatening |
| | QTc interval | QTc interval | QTc interval | consequences, |
| | 0.450 to 0.464 | 0.465 to 0.479 | ≥ 0.480 sec | eg, Torsade de |
| | sec | sec | | pointes or other |
| | | | | associated |
| | | | | serious |
| | | | | ventricular |
| | | | | dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein | Deep vein | Embolic event |
| | | thrombosis | thrombosis | (eg, pulmonary |
| | | AND No | AND | embolism, life- |
| | | intervention | Intervention | threatening |
| | | indicated (eg, | indicated (eg, | thrombus) |
| | | anticoagulation, | anticoagulation, | |
| | | lysis filter, | lysis filter, | |
| | | invasive | invasive | |
| | | procedure) | procedure) | |
| Vasovagal Episode | Present without | Present with | NA | NA |
| (associated with a | loss of | transient loss of | | |
| procedure of any kind) | consciousness | consciousness | | |

| CARDIOVASCULAR | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Ventricular | NA | Asymptomatic | New onset with | Life-threatening |
| Dysfunction | | diagnostic | symptoms OR | CHF |
| (congestive heart | | finding AND | Worsening | |
| failure, CHF) | | intervention | symptomatic | |
| | | indicated | CHF | |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm | FEV1 or peak | FEV1 or peak flow | FEV1 or peak | Cyanosis OR FEV1 |
| (acute) | flow reduced to | 50% to 69% | flow 25% to | or peak flow |
| | 70% to 80% | | 49% | < 25% OR |
| | | | | Intubation |
| Dyspnea or | Dyspnea on | Dyspnea on | Dyspnea at rest | Respiratory failure |
| Respiratory | exertion with no | exertion causing | causing inability | with ventilatory |
| Distress | or minimal | greater than | to perform | support indicated |
| | interference with | minimal | usual social & | |
| | usual social & | interference with | functional | |
| | functional | usual social & | activities | |
| | activities | functional | | |
| | | activities | | |
| Pediatric < 14 | Wheezing OR | Nasal flaring OR | Dyspnea at rest | Respiratory failure |
| Years | minimal increase | Intercostal | causing inability | with ventilatory |
| | in respiratory | retractions OR | to perform | support indicated |
| | rate for age | Pulse oximetry | usual social & | |
| | | 90% to 95% | functional | |
| | | | activities OR | |
| | | | Pulse oximetry | |
| | | | < 90% | |

| OCULAR/VISUAL | | | | |
|---------------|---------|---------|---------|---------|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |

| Uveitis | Asymptomatic | Symptomatic | Posterior or | Disabling visual |
|---|---|---|---|---|
| | but detectable on | anterior uveitis OR | pan-uveitis OR | loss in affected |
| | exam | Medical | Operative | eye(s) |
| | | intervention | intervention | |
| | | indicated | indicated | |
| Visual | Visual changes | Visual changes | Visual changes | Disabling visual |
| Changes | causing no or | causing greater | causing inability | loss in affected |
| (from | minimal | than minimal | to perform usual | eye(s) |
| baseline) | interference with | interference with | social & | |
| | usual social & | usual social & | functional | |
| | functional | functional | activities | |
| | activities | activities | | |

| SKIN | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |

| Cutaneous | Localized | Diffuse macular, | Diffuse macular, | Extensive or |
|---|---|---|---|---|
| Reaction – Rash | macular rash | maculopapular, | maculopapular, or | generalized |
| | | or morbilliform | morbilliform rash | bullous lesions |
| | | rash OR Target | with vesicles or | OR Stevens- |
| | | lesions | limited number of | Johnson |
| | | | bullae OR | syndrome OR |
| | | | Superficial | Ulceration of |
| | | | ulcerations of | mucous |
| | | | mucous | membrane |
| | | | membrane limited | involving two |
| | | | to one site | or more |
| | | | | distinct |
| | | | | mucosal sites |
| | | | | OR Toxic |
| | | | | epidermal |
| | | | | necrolysis |
| | | | | (TEN) |
| Hyperpigmentation | Slight or | Marked or | NA | NA |
| | localized | generalized | | |
| Hypopigmentation | Slight or | Marked or | NA | NA |
| | localized | generalized | | |
| Pruritis (itching – | Itching causing | Itching causing | Itching causing | NA |
| no skin lesions) | no or minimal | greater than | inability to | |
| | interference | minimal | perform usual | |
| (See also Injection | with usual | interference with | social & functional | |
| Site Reactions: | social & | usual social & | activities | |
| Pruritis associated | functional | functional | | |
| with injection) | activities | activities | | |

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of | Loss of appetite | Loss of appetite | Life- |
| | appetite | associated with | associated with | threatening |
| | without | decreased oral | significant weight | consequences |
| | decreased oral | intake without | loss | OR |
| | intake | significant weight | | Aggressive |
| | | loss | | intervention |
| | | | | indicated [eg, |
| | | | | tube feeding |
| | | | | or total |
| | | | | parenteral |
| | | | | nutrition] |
| Ascites | Asymptomatic | Symptomatic AND | Symptomatic | Life- |
| | | Intervention | despite | threatening |
| | | indicated (eg, | intervention | consequences |
| | | diuretics or | | |
| | | therapeutic | | |
| | | paracentesis) | | |
| Cholecystitis | NA | Symptomatic AND | Radiologic, | Life- |
| | | Medical | endoscopic, or | threatening |
| | | intervention | operative | consequences |
| | | indicated | intervention | (eg, sepsis or |
| | | | indicated | perforation) |
| Constipation | NA | Persistent | Obstipation with | Life- |
| | | constipation | manual evacuation | threatening |
| | | requiring regular | indicated | consequences |
| | | use of dietary | | (eg, |
| | | modifications, | | obstruction) |
| | | laxatives, or | | |
| | | enemas | | |

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Diarrhea | | | | |
| Adult and Pediatric | Transient or | Persistent | Bloody diarrhea | Life- |
| ≥ 1 Year | intermittent | episodes of | OR Increase of | threatening |
| | episodes of | unformed to | ≥ 7 stools per | consequences |
| | unformed | watery stools OR | 24-hour period OR | (eg, |
| | stools OR | Increase of 4-6 | IV fluid | hypotensive |
| | Increase of | stools over | replacement | shock) |
| | ≤ 3 stools over | baseline per | indicated | |
| | baseline/24 hr | 24 hrs. | | |
| Pediatric < 1 Year | Liquid stools | Liquid stools with | Liquid stools with | Liquid stools |
| | (more | increased number | moderate | resulting in |
| | unformed | of stools OR Mild | dehydration | severe |
| | than usual) | dehydration | | dehydration |
| | but usual | | | with |
| | number of | | | aggressive |
| | stools | | | rehydration |
| | | | | indicated OR |
| | | | | Hypotensive |
| | | | | shock |
| Dysphagia- | Symptomatic | Symptoms causing | Symptoms causing | Life- |
| Odynophagia | but able to eat | altered dietary | severely altered | threatening |
| | usual diet | intake without | dietary intake with | reduction in |
| | | medical | medical | oral intake |
| | | intervention | intervention | |
| | | indicated | indicated | |

| GASTROINTESTINAL | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucositis/Stomatitis | Erythema of | Patchy | Confluent | Tissue |
| (clinical exam) | the mucosa | pseudomembranes | pseudomembranes | necrosis OR |
| | | or ulcerations | or ulcerations OR | Diffuse |
| See also Proctitis, | | | Mucosal bleeding | spontaneous |
| Dysphagia- | | | with minor trauma | mucosal |
| Odynophagia | | | | bleeding OR |
| | | | | Life- |
| | | | | threatening |
| | | | | consequences |
| | | | | (eg, |
| | | | | aspiration, |
| | | | | choking) |
| Nausea | Transient | Persistent nausea | Persistent nausea | Life- |
| | (< 24 hours) | resulting in | resulting in | threatening |
| | or | decreased oral | minimal oral | consequences |
| | intermittent | intake for 24-48 | intake for > 48 | (eg, |
| | nausea with | hours | hours OR | hypotensive |
| | no or minimal | | Aggressive | shock) |
| | interference | | rehydration | |
| | with oral | | indicated (eg, | |
| | intake | | IV fluids) | |
| Pancreatitis | NA | Symptomatic AND | Symptomatic AND | Life- |
| | | Hospitalization not | Hospitalization | threatening |
| | | indicated (other | indicated (other | consequences |
| | | than ER visit) | than ER visit) | (eg, sepsis, |
| | | | | circulatory |
| | | | | failure, |
| | | | | hemorrhage) |

| GASTROINTESTINAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proctitis (functional- | Rectal | Symptoms causing | Symptoms causing | Life- |
| symptomatic) | discomfort | greater than | inability to | threatening |
| | AND No | minimal | perform usual | consequences |
| Also see Mucositis/ | intervention | interference with | social/ functional | (eg, |
| Stomatitis for | indicated | usual social & | activities OR | perforation) |
| Clinical Exam | | functional | Operative | |
| | | activities OR | intervention | |
| | | Medical | indicated | |
| | | intervention | | |
| | | indicated | | |
| Vomiting | Transient or | Frequent episodes | Persistent | Life- |
| | intermittent | of vomiting with | vomiting resulting | threatening |
| | vomiting with | no or mild | in orthostatic | consequences |
| | no or minimal | dehydration | hypotension OR | (eg, |
| | interference | | Aggressive | hypotensive |
| | with oral | | rehydration | shock) |
| | intake | | indicated | |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in | Alteration | Alteration | Alteration | Behavior |
| Personality-Behavior | causing no or | causing greater | causing | potentially |
| or in Mood (eg, | minimal | than minimal | inability to | harmful to self or |
| agitation, anxiety, | interference | interference | perform usual | others (eg, |
| depression, mania, | with usual | with usual social | social & | suicidal/homicidal |
| psychosis) | social & | & functional | functional | ideation or |
| | functional | activities | activities | attempt, acute |
| | activities | | | psychosis) OR |
| | | | | Causing inability |
| | | | | to perform basic |
| | | | | self-care functions |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Altered Mental Status | Changes | Mild lethargy or | Confusion, | Delirium OR |
| | causing no or | somnolence | memory | obtundation, OR |
| For Dementia, see | minimal | causing greater | impairment, | coma |
| Cognitive and | interference | than minimal | lethargy, or | |
| Behavioral/Attentiona | with usual | interference | somnolence | |
| l Disturbance | social & | with usual social | causing | |
| (including dementia | functional | & functional | inability to | |
| and ADD) | activities | activities | perform usual | |
| | | | social & | |
| | | | functional | |
| | | | activities | |
| Ataxia | Asymptomatic | Symptomatic | Symptomatic | Disabling ataxia |
| | ataxia | ataxia causing | ataxia causing | causing inability to |
| | detectable on | greater than | inability to | perform basic self- |
| | exam OR | minimal | perform usual | care functions |
| | Minimal | interference | social & | |
| | ataxia causing | with usual social | functional | |
| | no or minimal | & functional | activities | |
| | interference | activities | | |
| | with usual | | | |
| | social & | | | |
| | functional | | | |
| | activities | | | |
| Cognitive and | Disability | Disability | Disability | Disability causing |
| Behavioral/Attentiona | causing no or | causing greater | causing | inability to |
| l Disturbance | minimal | than minimal | inability to | perform basic self- |
| (including dementia | interference | interference | perform usual | care functions OR |
| and Attention Deficit | with usual | with usual social | social & | Institutionalizatio |
| Disorder) | social & | & functional | functional | n indicated |
| | functional | activities OR | activities OR | |
| | activities OR | Specialized | Specialized | |
| | Specialized | resources on | resources on a | |
| | resources not | part-time basis | full-time basis | |
| | indicated | indicated | indicated | |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| CNS Ischemia<br>(acute) | NA | NA | Transient<br>ischemic<br>attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |
| Developmental delay - | Mild | Moderate | Severe | Developmental |
| Pediatric ≤ 16 Years | developmenta | developmental | developmenta | regression, either |
| | l delay, either | delay, either | l delay, either | motor or |
| | motor or | motor or | motor or | cognitive, as |
| | cognitive, as | cognitive, as | cognitive, as | determined by |
| | determined by | determined by | determined by | comparison with a |
| | comparison | comparison | comparison | developmental |
| | with a | with a | with a | screening tool |
| | developmenta | developmental | developmenta | appropriate for |
| | l screening | screening tool | l screening | the setting |
| | tool | appropriate for | tool | |
| | appropriate | the setting | appropriate | |
| | for the setting | | for the setting | |
| Headache | Symptoms | Symptoms | Symptoms | Symptoms causing |
| | causing no or | causing greater | causing | inability to |
| | minimal | than minimal | inability to | perform basic self- |
| | interference | interference | perform usual | care functions OR |
| | with usual | with usual social | social & | Hospitalization |
| | social & | & functional | functional | indicated (other |
| | functional | activities | activities | than ER visit) OR |
| | activities | | | Headache with |
| | | | | significant |
| | | | | impairment of |
| | | | | alertness or other |
| | | | | neurologic |
| | | | | function |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Insomnia | NA | Difficulty | Difficulty | Disabling |
| | | sleeping causing | sleeping | insomnia causing |
| | | greater than | causing | inability to |
| | | minimal | inability to | perform basic self- |
| | | interference | perform usual | care functions |
| | | with usual | social & | |
| | | social/functiona | functional | |
| | | l activities | activities | |
| Neuromuscular | Asymptomatic | Muscle | Muscle | Disabling muscle |
| Weakness | with | weakness | weakness | weakness causing |
| (including myopathy & | decreased | causing greater | causing | inability to |
| neuropathy) | strength on | than minimal | inability to | perform basic self- |
| | exam OR | interference | perform usual | care functions OR |
| | Minimal | with usual social | social & | Respiratory |
| | muscle weak- | & functional | functional | muscle weakness |
| | ness causing | activities | activities | impairing |
| | no or minimal | | | ventilation |
| | interference | | | |
| | with usual | | | |
| | social & | | | |
| | functional | | | |
| | activities | | | |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Neurosensory | Asymptomatic | Sensory | Sensory | Disabling sensory |
| Alteration (including | with sensory | alteration or | alteration or | alteration or |
| paresthesia and | alteration on | paresthesia | paresthesia | paresthesia |
| painful neuropathy) | exam or | causing greater | causing | causing inability to |
| | minimal | than minimal | inability to | perform basic self- |
| | paresthesia | interference | perform usual | care functions |
| | causing no or | with usual social | social & | |
| | minimal | & functional | functional | |
| | interference | activities | activities | |
| | with usual | | | |
| | social & | | | |
| | functional | | | |
| | activities | | | |
| Seizure: (new onset) | NA | 1 seizure | 2-4 seizures | Seizures of any |
| | | | | kind that are |
| | | | | prolonged, |
| | | | | repetitive (eg, |
| | | | | status epilepticus), |
| | | | | or difficult to |
| | | | | control (eg, |
| | | | | refractory |
| | | | | epilepsy) |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Seizure: (pre-existing) | NA | Increased | Change in | Seizures of any |
| | | frequency of | seizure | kind that are |
| For Worsening of | | pre-existing | character | prolonged, |
| Existing Epilepsy the | | seizures (non- | from baseline | repetitive (eg, |
| Grades Should Be | | repetitive) | either in | status epilepticus), |
| Based on an Increase | | without change | duration or | or difficult to |
| from Previous Level of | | in seizure | quality (eg, | control (eg, |
| Control to Any of | | character OR | severity or | refractory |
| These Levels | | infrequent | focality) | epilepsy) |
| | | breakthrough | | |
| | | seizures while | | |
| | | on stable meds | | |
| | | in a previously | | |
| | | controlled | | |
| | | seizure disorder | | |
| Seizure | Seizure, | Seizure, | Seizure, | Seizure, |
| - Pediatric < 18 Years | generalized | generalized | generalized | generalized onset |
| | onset with or | onset with or | onset with or | with or without |
| | without | without | without | secondary |
| | secondary | secondary | secondary | generalization, |
| | generalization | generalization, | generalization | requiring |
| | , lasting | lasting 5–20 | , lasting | intubation and |
| | < 5 minutes | minutes with | > 20 minutes | sedation |
| | with | < 24 hours post | | |
| | < 24 hours | ictal state | | |
| | post ictal state | | | |
| Syncope (not | NA | Present | NA | NA |
| associated with a | | | | |
| procedure) | | | | |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Vertigo | Vertigo | Vertigo causing | Vertigo | Disabling vertigo |
| | causing no or | greater than | causing | causing inability to |
| | minimal | minimal | inability to | perform basic self- |
| | interference | interference | perform usual | care functions |
| | with usual | with usual social | social & | |
| | social & | & functional | functional | |
| | functional | activities | activities | |
| | activities | | | |

| MUSCULOSKEL | ETAL | | - | - |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia | Joint pain | Joint pain causing | Joint pain | Disabling joint |
| | causing no or | greater than | causing inability | pain causing |
| See also | minimal | minimal | to perform usual | inability to |
| Arthritis | interference | interference with | social & | perform basic |
| | with usual social | usual social & | functional | self-care |
| | & functional | functional activities | activities | functions |
| | activities | | | |
| Arthritis | Stiffness or joint | Stiffness or joint | Stiffness or joint | Disabling joint |
| | swelling causing | swelling causing | swelling causing | stiffness or |
| See also | no or minimal | greater than | inability to | swelling causing |
| Arthralgia | interference | minimal | perform usual | inability to |
| | with usual social | interference with | social & | perform basic |
| | & functional | usual social & | functional | self-care |
| | activities | functional activities | activities | functions |
| Bone Mineral | BMD t-score or | BMD t-score or z- | Pathological | Pathologic |
| Loss | z-score | score < -2.5 | fracture | fracture causing |
| | -2.5 to -1.0 | | (including loss | life-threatening |
| | | | of vertebral | consequences |
| | | | height) | |

| MUSCULOSKELETAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pediatric | BMD z-score | BMD z-score < -2.5 | Pathological | Pathologic |
| < 21 Years | −2.5 to −1.0 | | fracture | fracture causing |
| | | | (including loss | life-threatening |
| | | | of vertebral | consequences |
| | | | height) | |
| Myalgia | Muscle pain | Muscle pain causing | Muscle pain | Disabling muscle |
| (non-injection | causing no or | greater than | causing inability | pain causing |
| site) | minimal | minimal | to perform usual | inability to |
| | interference | interference with | social & | perform basic |
| | with usual social | usual social & | functional | self-care |
| | & functional | functional activities | activities | functions |
| | activities | | | |
| Osteonecrosis | NUCs | Asymptomatic with | Symptomatic | Disabling bone |
| | | radiographic | bone pain with | pain with |
| | | findings AND No | radiographic | radiographic |
| | | operative | findings OR | findings causing |
| | | intervention | Operative | inability to |
| | | indicated | intervention | perform basic |
| | | | indicated | self-care |
| | | | | functions |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Acute Systemic | Localized | Localized urticaria | Generalized | Acute anaphylaxis |
| Allergic | urticaria | with medical | urticaria OR | OR Life- |
| Reaction | (wheals) with | intervention | Angioedema with | threatening |
| | no medical | indicated OR Mild | medical | bronchospasm |
| | intervention | angioedema with no | intervention | OR laryngeal |
| | indicated | medical intervention | indicated OR | edema |
| | | indicated | Symptomatic | |
| | | | mild | |
| | | | bronchospasm | |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Chills | Symptoms | Symptoms causing | Symptoms | NA |
| | causing no or | greater than | causing inability | |
| | minimal | minimal | to perform usual | |
| | interference | interference with | social & | |
| | with usual | usual social & | functional | |
| | social & | functional activities | activities | |
| | functional | | | |
| | activities | | | |
| Fatigue | Symptoms | Symptoms causing | Symptoms | Incapacitating |
| | causing no or | greater than | causing inability | fatigue/malaise |
| Malaise | minimal | minimal | to perform usual | symptoms |
| | interference | interference with | social & | causing inability |
| | with usual | usual social & | functional | to perform basic |
| | social & | functional activities | activities | self-care |
| | functional | | | functions |
| | activities | | | |
| Fever | 37.7°C to | 38.7°C to 39.3°C | 39.4°C to 40.5°C | > 40.5°C |
| (nonaxillary) | 38.6°C | | | |
| | | 101.6°F to 102.8°F | 102.9°F to | > 104.9°F |
| | 99.8°F to | | 104.9°F | |
| | 101.5°F | | | |
| Pain- Indicate | Pain causing | Pain causing greater | Pain causing | Disabling pain |
| Body Site | no or minimal | than minimal | inability to | causing inability |
| | interference | interference with | perform usual | to perform basic |
| See also | with usual | usual social & | social & | self-care |
| Injection Site | social & | functional activities | functional | functions OR |
| Pain, | functional | | activities | Hospitalization |
| Headache, | activities | | | (other than ER |
| Arthralgia, and | | | | visit) indicated |
| Myalgia | | | | |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Unintentional | NA | 5% to 9% loss in | 10% to 19% loss | ≥ 20% loss in |
| Weight Loss | | body weight from | in body weight | body weight from |
| | | baseline | from baseline | baseline OR |
| | | | | Aggressive |
| | | | | intervention |
| | | | | indicated [eg, |
| | | | | tube feeding or |
| | | | | total parenteral |
| | | | | nutrition] |

| INJECTION SITE REACTION | | | | |
|---|---|---|---|---|
| · | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Injection Site | Pain/tenderness | Pain/tenderness | Pain/tenderness | Pain/tenderness |
| Pain (pain | causing no or | limiting use of | causing inability | causing inability to |
| without | minimal | limb OR | to perform usual | perform basic self- |
| touching) | limitation of use | Pain/tenderness | social & | care function OR |
| | of limb | causing greater | functional | Hospitalization |
| Or Tenderness | | than minimal | activities | (other than ER |
| (pain when area | | interference with | | visit) indicated for |
| is touched) | | usual social & | | management of |
| | | functional | | pain/tenderness |
| | | activities | | |
| Injection Site | Erythema OR | Erythema OR | Ulceration OR | Necrosis (involving |
| Reaction | Induration | Induration OR | Secondary | dermis and deeper |
| (Localized), | of $5 \times 5$ cm to | Edema > 9 cm any | infection OR | tissue) |
| > 15 Years | 9 × 9 cm (or | diameter (or > | Phlebitis OR | |
| | 25–81 × cm2) | 81 cm2) | Sterile abscess | |
| | | | OR Drainage | |
| Pediatric | Erythema OR | Erythema OR | Erythema OR | Necrosis (involving |
| ≤ 15 Years | Induration OR | Induration OR | Induration OR | dermis and deeper |
| | Edema present | Edema > 2.5 cm | Edema involving | tissue) |
| | but ≤ 2.5 cm | diameter but | ≥ 50% surface | |
| | diameter | < 50% surface | area of the | |
| | | area of the | extremity | |

| | | extremity | segment (eg, | |
|---|---|---|---|---|
| | | segment (eg, | upper | |
| | | upper arm/thigh) | arm/thigh) OR | |
| | | | Ulceration OR | |
| | | | Secondary | |
| | | | infection OR | |
| | | | Phlebitis OR | |
| | | | Sterile abscess | |
| | | | OR Drainage | |
| Pruritis | Itching localized | Itching beyond | Generalized | NA |
| Associated with | to injection site | the injection site | itching causing | |
| Injection | AND Relieved | but not | inability to | |
| | spontaneously | generalized OR | perform usual | |
| See also Skin: | or with < 48 h | Itching localized | social & | |
| Pruritis | treatment | to injection site | functional | |
| (itching—no | | requiring≥48 h | activities | |
| skin lesions) | | treatment | | |

| ENDOCRINE/METABOLIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy | Detectable by | Detectable on | Disfiguring OR | NA |
| (eg, back of neck, | study | physical exam by | Obvious changes | |
| breasts, | participant or | health care provider | on casual visual | |
| abdomen) | caregiver (for | | inspection | |
| | young | | | |
| | children and | | | |
| | disabled | | | |
| | adults) | | | |
| Diabetes | NA | New onset without | New onset with | Life-threatening |
| Mellitus | | need to initiate | initiation of | consequences |
| | | medication OR | indicated med | (eg, ketoacidosis, |
| | | Modification of | OR Diabetes | hyperosmolar |
| | | current meds to | uncontrolled | non-ketotic |
| | | regain glucose | despite | coma) |
| | | control | treatment | |
| | | | modification | |

| ENDOCRINE/METABOLIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Gynecomastia | Detectable by | Detectable on | Disfiguring OR | NA |
| | study | physical exam by | Obvious on | |
| | participant or | health care provider | casual visual | |
| | caregiver (for | | inspection | |
| | young | | | |
| | children and | | | |
| | disabled | | | |
| | adults) | | | |
| Hyperthyroidism | Asymptomatic | Symptomatic | Symptoms | Life-threatening |
| | | causing greater than | causing inability | consequences |
| | | minimal | to perform usual | (eg, thyroid |
| | | interference with | social & | storm) |
| | | usual social & | functional | |
| | | functional activities | activities OR | |
| | | OR Thyroid | Uncontrolled | |
| | | suppression | despite | |
| | | therapy indicated | treatment | |
| | | | modification | |
| Hypothyroidism | Asymptomatic | Symptomatic | Symptoms | Life-threatening |
| | | causing greater than | causing inability | consequences |
| | | minimal | to perform usual | (eg, myxedema |
| | | interference with | social & | coma) |
| | | usual social & | functional | |
| | | functional activities | activities OR | |
| | | OR Thyroid | Uncontrolled | |
| | | replacement | despite | |
| | | therapy indicated | treatment | |
| | | | modification | |

| ENDOCRINE/METABOLIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipoatrophy (eg, | Detectable by | Detectable on | Disfiguring OR | NA |
| fat loss from the | study | physical exam by | Obvious on | |
| face, extremities, | participant or | health care provider | casual visual | |
| buttocks) | caregiver (for | | inspection | |
| | young | | | |
| | children and | | | |
| | disabled | | | |
| | adults) | | | |

| GENITOURINUCsRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual | Spotting observed | Intermenstrual | Intermenstrual | Hemorrhage |
| Bleeding (IMB) | by participant OR | bleeding not | bleeding greater in | with life- |
| | Minimal blood | greater in | duration or | threatening |
| | observed during | duration or | amount than usual | hypotension OR |
| | clinical or | amount than | menstrual cycle | Operative |
| | colposcopic exam | usual menstrual | | intervention |
| | | cycle | | indicated |
| Urinary Tract | NA | Signs or | Signs or symptoms | Obstruction |
| obstruction | | symptoms of | of urinary tract | causing life- |
| (eg, stone) | | urinary tract | obstruction with | threatening |
| | | obstruction | hydronephrosis or | consequences |
| | | without | renal dysfunction | |
| | | hydronephrosis | | |
| | | or renal | | |
| | | dysfunction | | |

| INFECTION | | | | |
|-----------|---------|---------|---------|---------|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |

| Infection (any | Localized, no | Systemic | Systemic antiµbial | Life-threatening |
|---|---|---|---|---|
| other than | systemic antiµbial | antiµbial | treatment | consequences |
| HIV infection) | treatment | treatment | indicated AND | (eg, septic |
| | indicated AND | indicated OR | Symptoms causing | shock) |
| | Symptoms causing | Symptoms | inability to | |
| | no or minimal | causing greater | perform usual | |
| | interference with | than minimal | social & functional | |
| | usual social & | interference with | activities OR | |
| | functional | usual social & | Operative | |
| | activities | functional | intervention (other | |
| | | activities | than simple | |
| | | | incision and | |
| | | | drainage) indicated | |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement,
 continence, and feeding.

Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc